CLINICAL TRIAL: NCT01392378
Title: A Phase 4, Randomized, Open-Label Trial To Assess The Impact Of Prophylactic Antipyretic Medication On The Immunogenicity Of 13-Valent Pneumococcal Conjugate Vaccine Given With Routine Pediatric Vaccinations In Healthy Infants
Brief Title: Study Assessing the Effect of Medications to Prevent Fever on Prevenar 13®
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B1851047; 6096A1-4027
Record Dates: First submitted 2011-07-08; First posted 2011-07-12 (Estimated); Results first posted 2014-02-26 (Estimated); Last update posted 2014-02-26 (Estimated); Status verified 2014-01

CONDITIONS: Pneumococcal Vaccines
Keywords: Prevenar 13; 13vPnC; Antipyretic medication; Healthy subjects
MeSH Terms: interventions — diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine; Acetaminophen; Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group 1 (Experimental): Subjects will receive 13-valent pneumococcal vaccine and INFANRIX hexa at 2, 3, 4 and 12 months of age. They will also receive 2 doses of paracetamol on the day of each vaccination.
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine; Biological: INFANRIX hexa; Drug: Paracetamol
- Group 2 (Experimental): Subjects will receive 13-valent pneumococcal vaccine and INFANRIX hexa at 2, 3, 4 and 12 months of age. They will also receive 2 doses of ibuprofen on the day of each vaccination.the first dose.
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine; Biological: INFANRIX hexa; Drug: Ibuprofen
- Group 3 (Experimental): Subjects will receive 13-valent pneumococcal vaccine and INFANRIX hexa at 2, 3, 4 and 12 months of age. They will also receive 3 doses of paracetamol on the day of each vaccination.
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine; Biological: INFANRIX hexa; Drug: Paracetamol
- Group 4 (Experimental): Subjects will receive 13-valent pneumococcal vaccine and INFANRIX hexa at 2, 3, 4 and 12 months of age. They will also receive 3 doses of ibuprofen on the day of each vaccination.
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine; Biological: INFANRIX hexa; Drug: Ibuprofen
- Group 5 (Experimental): Subjects will receive 13-valent pneumococcal vaccine and INFANRIX hexa at 2, 3, 4 and 12 months of age. This group does not receive any antipyretic medication as part of the study.
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine; Biological: INFANRIX hexa

INTERVENTIONS:
Biological: 13-valent pneumococcal conjugate vaccine — 13vPnC will be administered by intramuscular injection at 2, 3, 4 and 12 months of age.
  Arms: Group 1
Biological: INFANRIX hexa — INFANRIX hexa will be administered by intramuscular injection at 2, 3, 4 and 12 months of age.
  Arms: Group 1
Drug: Paracetamol — Paracetamol suspension for oral administration will be given at a weight adjusted dose of 15mg/kg/dose. The first dose will be given 6-8 hours after each vaccination, the second dose to be given 6-8 hours after the first.
  Arms: Group 1
Biological: 13-valent pneumococcal conjugate vaccine — 13vPnC will be administered by intramuscular injection at 2, 3, 4 and 12 months of age.
  Arms: Group 2
Biological: INFANRIX hexa — INFANRIX hexa will be administered by intramuscular injection at 2, 3, 4 and 12 months of age.
  Arms: Group 2
Drug: Ibuprofen — Ibuprofen suspension for oral administration will be given at a weight adjusted dose of 10mg/kg/dose. The first dose will be given 6-8 hours after each vaccination, the second dose to be given 6-8 hours after the first.
  Arms: Group 2
Biological: 13-valent pneumococcal conjugate vaccine — 13vPnC will be administered by intramuscular injection at 2, 3, 4 and 12 months of age.
  Arms: Group 3
Biological: INFANRIX hexa — INFANRIX hexa will be administered by intramuscular injection at 2, 3, 4 and 12 months of age.
  Arms: Group 3
Drug: Paracetamol — Paracetamol suspension for oral administration will be given at a weight adjusted dose of 15mg/kg/dose. The first dose will be given at the time of each vaccination, the second dose to be given 6-8 hours after the first, and the third dose to be given 6-8 hours after the second.
  Arms: Group 3
Biological: 13-valent pneumococcal conjugate vaccine — 13vPnC will be administered by intramuscular injection at 2, 3, 4 and 12 months of age.
  Arms: Group 4
Biological: INFANRIX hexa — INFANRIX hexa will be administered by intramuscular injection at 2, 3, 4 and 12 months of age.
  Arms: Group 4
Drug: Ibuprofen — Ibuprofen suspension for oral administration will be given at a weight adjusted dose of 10mg/kg/dose. The first dose will be given at the time of each vaccination, the second dose to be given 6-8 hours after the first, and the third dose to be given 6-8 hours after the second.
  Arms: Group 4
Biological: 13-valent pneumococcal conjugate vaccine — 13vPnC will be administered by intramuscular injection at 2, 3, 4 and 12 months of age.
  Arms: Group 5
Biological: INFANRIX hexa — INFANRIX hexa will be administered by intramuscular injection at 2, 3, 4 and 12 months of age.
  Arms: Group 5

SUMMARY:
The purposes of this study are assess the immunological response (measure the amount of antibodies, i.e. proteins that fight off germs) produced by children after they have been given the 13-valent pneumococcal vaccine (13vPnC) and INFANRIX hexa at 2, 3, 4 and 12 months of age when medications to prevent fever are given on the same day as the vaccination. Also to evaluate the safety of 13-valent pneumococcal conjugate vaccine (13vPnC) in children who receive medications to prevent fever on the day of vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Aged 2 months (56 to 98 days) at time of enrollment.
* Healthy infant as determined by medical history, physical examination, and judgment of the investigator.

Exclusion Criteria:

* Previous vaccination with licensed or investigational pneumococcal, diphtheria, tetanus, pertussis, polio, or Hib conjugate vaccines.
* A previous anaphylactic reaction to any vaccine or vaccine-related component.
* Allergy or contraindication to paracetamol or ibuprofen administration.
* Contraindication to vaccination with pneumococcal conjugate, diphtheria, tetanus, pertussis, polio, Hib, or HBV vaccines.

Ages: 56 Days to 98 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 908 (Actual)
Dates: Start 2011-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (14):
- Poland (14):
  - Gabinet Lekarski, Dębica
  - Hanna Czajka Indywidualna Praktyka Lekarska, Krakow
  - NZOZ "Praktimed" sp. z o.o., Krakow
  - Specjalistyczna Praktyka Lekarska Gravita, Lodz
  - SP ZOZ Lubartow, Lubartów
  - NZOZ Praktyka Lekarza Rodzinnego Eskulap, Lublin
  - NZOZ Praktyka Lekarza Rodzinnego Alina Grocka-Wlazlak, Oborniki Śląskie
  - Specjalistyczny ZOZ nad Matka i Dzieckiem, Oddzial Obserwacyjno Zakazny A, Szpital Dzieciecy, Poznan
  - NZLA Michalkowice Jarosz i Partnerzy, Siemianowice Śląskie
  - NZOZ Nasz Lekarz, Torun
  - Szpital im. Sw. Jadwigi Slaskiej, Oddzia Pediatryczny, Trzebnica
  - DEN-MED Gabinet Lekarsko-Stomatologiczny Joanna i Jacek Witwiccy, Warsaw
  - Samodzielny Publiczny Szpital Kliniczny nr 1 we Wroclawiu, Wroclaw
  - NZOZ Salmed, Łęczna

REFERENCES:
- [Derived] Wysocki J, Center KJ, Brzostek J, Majda-Stanislawska E, Szymanski H, Szenborn L, Czajka H, Hasiec B, Dziduch J, Jackowska T, Witor A, Kopinska E, Konior R, Giardina PC, Sundaraiyer V, Patterson S, Gruber WC, Scott DA, Gurtman A. A randomized study of fever prophylaxis and the immunogenicity of routine pediatric vaccinations. Vaccine. 2017 Apr 4;35(15):1926-1935. doi: 10.1016/j.vaccine.2017.02.035. Epub 2017 Mar 3. PMID 28262330
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1851047&StudyName=Study%20Assessing%20the%20Effect%20of%20Medications%20to%20Prevent%20Fever%20on%20Prevenar%2013%AE

RESULTS

PARTICIPANT FLOW:
Groups:
- 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily: Participants received open-label 0.5 milliliter (mL) dose of 13-valent pneumococcal conjugate vaccine (13vPnC) intramuscularly and INFANRIX hexa intramuscularly as per manufacturer's instructions at 2 months (greater than or equal to [>=]56 to less than or equal to [<=]98 days of age), 3 months (28 to 42 days after Dose 1), 4 months (28 to 42 days after Dose 2, infant series) and 11 to 12 months (366 to 425 days of age, toddler dose) of age, along with paracetamol suspension 15 milligram per kilogram (mg/kg) orally at 6 to 8 hours after each vaccination and 6 to 8 hours after first dose of paracetamol.
- 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily: Participants received open-label 0.5 mL dose of 13vPnC intramuscularly and INFANRIX hexa intramuscularly as per manufacturer's instructions at 2 months (>=56 to <=98 days of age), 3 months (28 to 42 days after Dose 1), 4 months (28 to 42 days after Dose 2, infant series) and 11 to 12 months (366 to 425 days of age, toddler dose) of age, along with ibuprofen suspension 10 mg/kg orally at 6 to 8 hours after each vaccination and 6 to 8 hours after first dose of ibuprofen.
- 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily: Participants received open-label 0.5 mL dose of 13vPnC intramuscularly and INFANRIX hexa intramuscularly as per manufacturer's instructions at 2 months (>=56 to <=98 days of age), 3 months (28 to 42 days after Dose 1), 4 months (28 to 42 days after Dose 2, infant series) and 11 to 12 months (366 to 425 days of age, toddler dose) of age, along with paracetamol suspension 15 mg/kg orally immediately after vaccination, 6 to 8 hours after vaccination and 6 to 8 hours after last dose of paracetamol.
- 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily: Participants received open-label 0.5 mL dose of 13vPnC intramuscularly and INFANRIX hexa intramuscularly as per manufacturer's instructions at 2 months (>=56 to <=98 days of age), 3 months (28 to 42 days after Dose 1), 4 months (28 to 42 days after Dose 2, infant series) and 11 to 12 months (366 to 425 days of age, toddler dose) of age, along with ibuprofen suspension 10 mg/kg orally immediately after vaccination, 6 to 8 hours after vaccination and 6 to 8 hours after last dose of ibuprofen.
- 13vPnC + INFANRIX Hexa: Participants received open-label 0.5 mL dose of 13vPnC intramuscularly and INFANRIX hexa intramuscularly as per manufacturer's instructions at 2 months (>=56 to <=98 days of age), 3 months (28 to 42 days after Dose 1), 4 months (28 to 42 days after Dose 2, infant series) and 11 to 12 months (366 to 425 days of age, toddler dose) of age.
Period: Infant Series
Arm/Group | 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily | 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily | 13vPnC + INFANRIX Hexa
Started | 173 | 176 | 172 | 177 | 210
Vaccinated Dose 1 | 173 | 176 | 172 | 177 | 210
Vaccinated Dose 2 | 171 | 174 | 172 | 177 | 210
Vaccinated Dose 3 | 170 | 174 | 172 | 176 | 210
Completed | 169 | 174 | 172 | 175 | 210
Not Completed | 4 | 2 | 0 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Parent | 4 | 1 | 0 | 0 | 0
Period: After Infant Series
Arm/Group | 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily | 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily | 13vPnC + INFANRIX Hexa
Started | 169 | 174 | 172 | 175 | 210
Completed | 169 | 173 | 170 | 175 | 209
Not Completed | 0 | 1 | 2 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Parent | 0 | 1 | 1 | 0 | 1
Period: Toddler Dose
Arm/Group | 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily | 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily | 13vPnC + INFANRIX Hexa
Started | 169 | 173 | 170 | 175 | 209
Completed | 169 | 172 | 170 | 173 | 208
Not Completed | 0 | 1 | 0 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Parent | 0 | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily | 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily | 13vPnC + INFANRIX Hexa | Total
Number analyzed (Participants) | 173 | 176 | 172 | 177 | 210 | 908
Age, Continuous [Mean (Standard Deviation); unit: days] | 65.1 (9.5) | 66.5 (10.1) | 65.6 (9.7) | 66.4 (10.3) | 65.6 (9.4) | 65.8 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 89 | 75 | 79 | 98 | 428
  Male | 86 | 87 | 97 | 98 | 112 | 480

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Concentration (GMC) for Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody 1 Month After the Infant Series
Description: Antibody geometric least squares (LS) mean concentrations (GMCs) for 13 pneumococcal serotypes (4, 6B, 9V, 14, 18C, 19F, 23F, 1, 3, 5, 6A, 7F and 19A) are presented. GMC (13vPnC) and corresponding 2-sided 95 percent (%) confidence interval (CI) were evaluated. Geometric means (GMs) were calculated using all participants with available data for the specified blood draw. Here 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure and 'n' signifies participants with a determinate IgG concentration to the given serotype for each arm, respectively.
Time Frame: 1 month after the infant series
Population: Modified intent-to-treat (mITT) infant immunogenicity set: all eligible participants who had >=1 valid,determinate assay result, 56-98 days of age at Vaccination 1, received antipyretic regimen as per randomization,may have had received additional anti-pyretic medication,had blood drawn within specified time frames,had no major protocol violations.
Measure: Geometric Mean (95% Confidence Interval); unit: microgram per milliliter (mcg/mL)
Arm/Group | 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily | 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily | 13vPnC + INFANRIX Hexa
Number analyzed (Participants) | 138 | 155 | 148 | 147 | 210
microgram per milliliter (mcg/mL)
  4 (n = 137, 155, 148, 146, 210) | 1.64 [1.44 to 1.87] | 1.99 [1.76 to 2.25] | 1.48 [1.31 to 1.68] | 2.07 [1.82 to 2.34] | 2.02 [1.82 to 2.25]
  6B (n = 136, 155, 148, 146, 210) | 0.68 [0.55 to 0.83] | 0.91 [0.76 to 1.10] | 0.56 [0.46 to 0.68] | 0.90 [0.74 to 1.09] | 0.81 [0.69 to 0.96]
  9V (n = 138, 155, 148, 147, 210) | 1.13 [1.01 to 1.27] | 1.45 [1.30 to 1.61] | 1.17 [1.05 to 1.30] | 1.40 [1.26 to 1.56] | 1.31 [1.19 to 1.43]
  14 (n = 138, 155, 148, 147, 210) | 4.45 [3.76 to 5.26] | 4.73 [4.04 to 5.54] | 4.75 [4.04 to 5.58] | 5.26 [4.48 to 6.19] | 5.38 [4.70 to 6.16]
  18C (n = 138, 155, 148, 147, 210) | 1.47 [1.29 to 1.66] | 1.73 [1.54 to 1.95] | 1.25 [1.11 to 1.42] | 1.75 [1.55 to 1.97] | 1.54 [1.39 to 1.70]
  19F (n = 138, 155, 148, 147, 210) | 1.78 [1.57 to 2.02] | 2.30 [2.04 to 2.59] | 1.59 [1.41 to 1.80] | 2.04 [1.81 to 2.31] | 1.99 [1.80 to 2.20]
  23F (n= 137, 155, 148, 146, 210) | 0.85 [0.72 to 1.00] | 1.19 [1.02 to 1.40] | 0.73 [0.62 to 0.86] | 1.07 [0.91 to 1.26] | 1.04 [0.91 to 1.19]
  1 (n = 138, 155, 148, 147, 210) | 1.12 [0.98 to 1.27] | 1.50 [1.33 to 1.69] | 1.02 [0.90 to 1.16] | 1.29 [1.14 to 1.47] | 1.25 [1.12 to 1.38]
  3 (n = 138, 155, 148, 147, 210) | 0.71 [0.63 to 0.79] | 0.83 [0.75 to 0.93] | 0.57 [0.51 to 0.64] | 0.84 [0.75 to 0.94] | 0.88 [0.79 to 0.96]
  5 (n = 137, 155, 148, 146, 210) | 0.79 [0.69 to 0.91] | 0.98 [0.86 to 1.11] | 0.63 [0.55 to 0.72] | 0.90 [0.78 to 1.02] | 0.81 [0.73 to 0.91]
  6A (n = 138, 155, 148, 146, 210) | 0.97 [0.84 to 1.13] | 1.25 [1.09 to 1.44] | 0.85 [0.74 to 0.98] | 1.22 [1.06 to 1.41] | 1.10 [0.97 to 1.24]
  7F (n = 138, 155, 148, 146, 210) | 1.94 [1.74 to 2.16] | 2.22 [2.01 to 2.46] | 1.83 [1.65 to 2.03] | 2.28 [2.06 to 2.53] | 2.15 [1.97 to 2.34]
  19A (n = 137, 155, 148, 146, 210) | 2.70 [2.38 to 3.07] | 3.39 [3.01 to 3.82] | 2.53 [2.24 to 2.86] | 3.14 [2.77 to 3.55] | 3.02 [2.72 to 3.34]
Statistical Analysis 1: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 4: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.0856, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.81, 95% CI 2-sided [0.69 to 0.96]
Statistical Analysis 2: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 4: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.8546, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.99, 95% CI 2-sided [0.84 to 1.16]
Statistical Analysis 3: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 4: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.0012, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.73, 95% CI 2-sided [0.62 to 0.86]
Statistical Analysis 4: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 4: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.8414, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.02, 95% CI 2-sided [0.87 to 1.20]
Statistical Analysis 5: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 6B: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.2412, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.83, 95% CI 2-sided [0.64 to 1.08]
Statistical Analysis 6: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 6B: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.4548, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.13, 95% CI 2-sided [0.88 to 1.44]
Statistical Analysis 7: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 6B: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.0093, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.69, 95% CI 2-sided [0.53 to 0.88]
Statistical Analysis 8: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 6B: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.8414, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.10, 95% CI 2-sided [0.86 to 1.42]
Statistical Analysis 9: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 9V: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.1749, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.87, 95% CI 2-sided [0.75 to 1.00]
Statistical Analysis 10: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 9V: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.3121, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.11, 95% CI 2-sided [0.96 to 1.27]
Statistical Analysis 11: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 9V: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.1351, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.89, 95% CI 2-sided [0.78 to 1.03]
Statistical Analysis 12: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 9V: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.8414, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.07, 95% CI 2-sided [0.93 to 1.24]
Statistical Analysis 13: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 14: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.2158, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.83, 95% CI 2-sided [0.67 to 1.03]
Statistical Analysis 14: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 14: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.3279, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.88, 95% CI 2-sided [0.71 to 1.08]
Statistical Analysis 15: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 14: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.2472, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.88, 95% CI 2-sided [0.72 to 1.09]
Statistical Analysis 16: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 14: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.8414, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.98, 95% CI 2-sided [0.79 to 1.21]
Statistical Analysis 17: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 18C: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.6193, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.95, 95% CI 2-sided [0.81 to 1.12]
Statistical Analysis 18: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 18C: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.3121, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.13, 95% CI 2-sided [0.96 to 1.32]
Statistical Analysis 19: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 18C: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.0191, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.82, 95% CI 2-sided [0.70 to 0.96]
Statistical Analysis 20: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 18C: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.8414, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.14, 95% CI 2-sided [0.97 to 1.33]
Statistical Analysis 21: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 19F: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.2412, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.90, 95% CI 2-sided [0.76 to 1.05]
Statistical Analysis 22: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 19F: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.3121, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.15, 95% CI 2-sided [0.99 to 1.35]
Statistical Analysis 23: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 19F: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.0135, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.80, 95% CI 2-sided [0.68 to 0.94]
Statistical Analysis 24: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 19F: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.8414, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.03, 95% CI 2-sided [0.87 to 1.21]
Statistical Analysis 25: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 23F: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.1749, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.81, 95% CI 2-sided [0.66 to 1.00]
Statistical Analysis 26: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 23F: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.3121, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.15, 95% CI 2-sided [0.93 to 1.41]
Statistical Analysis 27: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 23F: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.0038, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.70, 95% CI 2-sided [0.57 to 0.86]
Statistical Analysis 28: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 23F: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.8414, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.03, 95% CI 2-sided [0.84 to 1.27]
Statistical Analysis 29: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 1: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.2412, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.90, 95% CI 2-sided [0.76 to 1.06]
Statistical Analysis 30: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 1: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.2053, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.20, 95% CI 2-sided [1.02 to 1.41]
Statistical Analysis 31: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 1: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.0241, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.82, 95% CI 2-sided [0.70 to 0.96]
Statistical Analysis 32: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 1: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.8414, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.04, 95% CI 2-sided [0.88 to 1.22]
Statistical Analysis 33: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 3: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.0732, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.81, 95% CI 2-sided [0.69 to 0.94]
Statistical Analysis 34: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 3: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.6090, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.95, 95% CI 2-sided [0.82 to 1.10]
Statistical Analysis 35: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 3: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p < 0.0001, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.65, 95% CI 2-sided [0.56 to 0.76]
Statistical Analysis 36: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 3: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.8414, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.96, 95% CI 2-sided [0.82 to 1.11]
Statistical Analysis 37: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 5: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.7828, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.98, 95% CI 2-sided [0.82 to 1.16]
Statistical Analysis 38: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 5: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.2053, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.21, 95% CI 2-sided [1.02 to 1.43]
Statistical Analysis 39: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 5: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.0093, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.77, 95% CI 2-sided [0.65 to 0.92]
Statistical Analysis 40: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 5: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.8414, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.11, 95% CI 2-sided [0.93 to 1.31]
Statistical Analysis 41: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 6A: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.2412, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.88, 95% CI 2-sided [0.73 to 1.07]
Statistical Analysis 42: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 6A: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.3121, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.14, 95% CI 2-sided [0.95 to 1.37]
Statistical Analysis 43: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 6A: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.0135, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.77, 95% CI 2-sided [0.64 to 0.93]
Statistical Analysis 44: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 6A: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.8414, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.11, 95% CI 2-sided [0.92 to 1.34]
Statistical Analysis 45: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 7F: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.2412, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.90, 95% CI 2-sided [0.79 to 1.03]
Statistical Analysis 46: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 7F: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.6652, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.03, 95% CI 2-sided [0.91 to 1.18]
Statistical Analysis 47: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 7F: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.0275, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.85, 95% CI 2-sided [0.75 to 0.98]
Statistical Analysis 48: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 7F: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.8414, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.06, 95% CI 2-sided [0.93 to 1.21]
Statistical Analysis 49: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 19A: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.2412, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.90, 95% CI 2-sided [0.76 to 1.06]
Statistical Analysis 50: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 19A: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.3121, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.13, 95% CI 2-sided [0.96 to 1.32]
Statistical Analysis 51: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 19A: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.0387, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.84, 95% CI 2-sided [0.72 to 0.99]
Statistical Analysis 52: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 19A: Ratio of IgG GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.8414, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.04, 95% CI 2-sided [0.89 to 1.22]

2. Secondary Outcome: Percentage of Participants Achieving Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody Level Greater Than or Equal to (>=)0.35 Microgram Per Milliliter (Mcg/mL) 1 Month After the Infant Series
Description: Percentage of participants achieving predefined antibody threshold >=0.35 mcg/mL along with the corresponding 95% confidence interval (CI) for 13 pneumococcal serotypes (4, 6B, 9V, 14, 18C, 19F, 23F, 1, 3, 5, 6A, 7F and 19A) are presented. Exact 2-sided CI based on the observed proportion of participants.
Time Frame: 1 month after the infant series
Population: mITT infant immunogenicity population. Here 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure and 'n' signifies participants with a determinate IgG concentration to the given serotype for each arm, respectively.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily | 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily | 13vPnC + INFANRIX Hexa
Number analyzed (Participants) | 138 | 155 | 148 | 147 | 210
percentage of participants
  4 (n = 137, 155, 148, 146, 210) | 96.4 [91.69 to 98.80] | 97.4 [93.52 to 99.29] | 96.6 [92.29 to 98.89] | 97.3 [93.13 to 99.25] | 98.1 [95.20 to 99.48]
  6B (n = 136, 155, 148, 146, 210) | 72.8 [64.50 to 80.07] | 80.0 [72.83 to 85.99] | 61.5 [53.14 to 69.36] | 79.5 [71.98 to 85.69] | 77.6 [71.37 to 83.07]
  9V (n = 138, 155, 148, 147, 210) | 94.2 [88.90 to 97.46] | 99.4 [96.46 to 99.98] | 95.9 [91.39 to 98.50] | 95.9 [91.33 to 98.49] | 96.2 [92.63 to 98.34]
  14 (n = 138, 155, 148, 147, 210) | 100.0 [97.36 to 100.00] | 98.7 [95.42 to 99.84] | 99.3 [96.29 to 99.98] | 98.6 [95.17 to 99.83] | 99.5 [97.38 to 99.99]
  18C (n = 138, 155, 148, 147, 210) | 96.4 [91.75 to 98.81] | 97.4 [93.52 to 99.29] | 95.3 [90.50 to 98.08] | 95.9 [91.33 to 98.49] | 96.7 [93.25 to 98.65]
  19F (n = 138, 155, 148, 147, 210) | 97.1 [92.74 to 99.20] | 99.4 [96.46 to 99.98] | 95.3 [90.50 to 98.08] | 96.6 [92.24 to 98.89] | 97.6 [94.53 to 99.22]
  23F (n = 137, 155, 148, 146, 210) | 86.1 [79.19 to 91.44] | 90.3 [84.54 to 94.48] | 74.3 [66.50 to 81.15] | 88.4 [82.01 to 93.07] | 88.1 [82.93 to 92.15]
  1 (n = 138, 155, 148, 147, 210) | 94.2 [88.90 to 97.46] | 97.4 [93.52 to 99.29] | 90.5 [84.64 to 94.73] | 94.6 [89.56 to 97.62] | 94.3 [90.23 to 97.01]
  3 (n = 138, 155, 148, 147, 210) | 83.3 [76.05 to 89.13] | 89.7 [83.78 to 93.98] | 81.1 [73.83 to 87.05] | 88.4 [82.13 to 93.12] | 91.0 [86.23 to 94.46]
  5 (n = 137, 155, 148, 146, 210) | 84.7 [77.53 to 90.25] | 91.0 [85.31 to 94.97] | 76.4 [68.68 to 82.94] | 89.7 [83.62 to 94.13] | 84.3 [78.65 to 88.93]
  6A (n = 138, 155, 148, 146, 210) | 86.2 [79.34 to 91.50] | 92.3 [86.87 to 95.94] | 83.1 [76.08 to 88.76] | 91.8 [86.08 to 95.68] | 91.9 [87.36 to 95.21]
  7F (n = 138, 155, 148, 146, 210) | 100.0 [97.36 to 100.00] | 99.4 [96.46 to 99.98] | 97.3 [93.22 to 99.26] | 100.0 [97.51 to 100.00] | 99.5 [97.38 to 99.99]
  19A (n = 137, 155, 148, 146, 210) | 98.5 [94.83 to 99.82] | 99.4 [96.46 to 99.98] | 98.0 [94.19 to 99.58] | 99.3 [96.24 to 99.98] | 100.0 [98.26 to 100.00]

3. Secondary Outcome: Geometric Mean Concentration (GMC) for Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody 1 Month After the Toddler Dose
Description: Antibody geometric LS mean concentrations (GMCs) for 13 pneumococcal serotypes (4, 6B, 9V, 14, 18C, 19F, 23F, 1, 3, 5, 6A, 7F and 19A) are presented. GMC (13vPnC) and corresponding 2-sided 95% CI were evaluated. Geometric means (GMs) were calculated using all participants with available data for the specified blood draw. Here 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure and 'n' signifies participants with a determinate IgG concentration to the given serotype for each arm respectively.
Time Frame: 1 month after the toddler dose
Population: mITT toddler immunogenicity set: eligible participants who had >=1 valid,determinate assay result, 56-98 days of age at Vaccination 1, received antipyretic regimen as per randomization, received all vaccinations, may have had received additional anti-pyretic medication, had blood drawn within specified time frames, had no major protocol violations.
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily | 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily | 13vPnC + INFANRIX Hexa
Number analyzed (Participants) | 130 | 144 | 143 | 139 | 206
mcg/mL
  4 (n = 130, 144, 143, 139, 206) | 3.07 [2.66 to 3.54] | 3.43 [3.00 to 3.93] | 2.97 [2.60 to 3.41] | 3.43 [2.99 to 3.94] | 3.10 [2.77 to 3.48]
  6B (n = 130, 144, 143, 139, 206) | 6.70 [5.76 to 7.78] | 8.01 [6.94 to 9.24] | 6.38 [5.53 to 7.36] | 7.30 [6.31 to 8.44] | 7.08 [6.28 to 7.98]
  9V (n = 130, 144, 143, 139, 206) | 2.15 [1.93 to 2.40] | 2.23 [2.01 to 2.47] | 2.17 [1.96 to 2.41] | 2.12 [1.91 to 2.35] | 2.16 [1.99 to 2.36]
  14 (n = 130, 144, 143, 139, 206) | 8.10 [7.04 to 9.31] | 8.40 [7.36 to 9.59] | 7.95 [6.96 to 9.08] | 9.12 [7.96 to 10.43] | 9.10 [8.15 to 10.17]
  18C (n = 130, 144, 143, 139, 206) | 1.35 [1.20 to 1.53] | 1.68 [1.49 to 1.88] | 1.36 [1.21 to 1.53] | 1.63 [1.45 to 1.84] | 1.59 [1.44 to 1.75]
  19F (n = 130, 144, 143, 139, 206) | 8.41 [7.17 to 9.87] | 8.99 [7.72 to 10.46] | 7.53 [6.47 to 8.76] | 8.02 [6.88 to 9.36] | 7.95 [7.00 to 9.02]
  23F (n = 130, 144, 142, 139, 206) | 2.34 [2.01 to 2.73] | 2.96 [2.56 to 3.43] | 2.37 [2.05 to 2.75] | 2.86 [2.47 to 3.32] | 2.75 [2.43 to 3.10]
  1 (n = 130, 144, 143, 139, 206) | 2.80 [2.47 to 3.17] | 3.22 [2.85 to 3.62] | 2.66 [2.36 to 3.00] | 3.12 [2.76 to 3.52] | 3.04 [2.75 to 3.35]
  3 (n = 129, 144, 143, 138, 203) | 0.46 [0.40 to 0.52] | 0.54 [0.47 to 0.61] | 0.46 [0.40 to 0.52] | 0.49 [0.42 to 0.55] | 0.54 [0.48 to 0.60]
  5 (n = 130, 144, 143, 139, 206) | 2.33 [2.07 to 2.63] | 2.75 [2.46 to 3.07] | 2.40 [2.15 to 2.69] | 2.62 [2.33 to 2.93] | 2.84 [2.59 to 3.12]
  6A (n = 130, 144, 143, 139, 206) | 5.12 [4.48 to 5.86] | 5.73 [5.04 to 6.50] | 5.27 [4.64 to 5.99] | 5.36 [4.70 to 6.10] | 5.52 [4.97 to 6.14]
  7F (n = 130, 144, 142, 139, 206) | 3.79 [3.42 to 4.19] | 3.89 [3.54 to 4.28] | 3.56 [3.23 to 3.92] | 3.97 [3.60 to 4.38] | 3.98 [3.67 to 4.31]
  19A (n = 129, 144, 142, 139, 206) | 7.11 [6.22 to 8.12] | 7.99 [7.04 to 9.06] | 7.31 [6.43 to 8.30] | 7.35 [6.47 to 8.36] | 7.71 [6.94 to 8.57]
Statistical Analysis 1: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9350, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.99, 95% CI 2-sided [0.82 to 1.19]
Statistical Analysis 2: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.7918, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.11, 95% CI 2-sided [0.93 to 1.32]
Statistical Analysis 3: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.6922, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.96, 95% CI 2-sided [0.80 to 1.14]
Statistical Analysis 4: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; p = 0.9765, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.11, 95% CI 2-sided [0.93 to 1.32]
Statistical Analysis 5: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; p = 0.6915, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.95, 95% CI 2-sided [0.78 to 1.15]
Statistical Analysis 6: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 6]; Test type: Superiority or Other; p = 0.7918, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.13, 95% CI 2-sided [0.94 to 1.36]
Statistical Analysis 7: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 7]; Test type: Superiority or Other; p = 0.4389, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.90, 95% CI 2-sided [0.75 to 1.09]
Statistical Analysis 8: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 8]; Test type: Superiority or Other; p = 0.9765, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.03, 95% CI 2-sided [0.85 to 1.24]
Statistical Analysis 9: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 9]; Test type: Superiority or Other; p = 0.9350, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.99, 95% CI 2-sided [0.87 to 1.14]
Statistical Analysis 10: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 10]; Test type: Superiority or Other; p = 0.7918, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.03, 95% CI 2-sided [0.90 to 1.18]
Statistical Analysis 11: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 11]; Test type: Superiority or Other; p = 0.9430, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.00, 95% CI 2-sided [0.88 to 1.15]
Statistical Analysis 12: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; p = 0.9765, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.98, 95% CI 2-sided [0.85 to 1.12]
Statistical Analysis 13: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 13]; Test type: Superiority or Other; p = 0.5167, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.89, 95% CI 2-sided [0.74 to 1.06]
Statistical Analysis 14: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 14]; Test type: Superiority or Other; p = 0.7918, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.92, 95% CI 2-sided [0.78 to 1.10]
Statistical Analysis 15: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 15]; Test type: Superiority or Other; p = 0.2514, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.87, 95% CI 2-sided [0.73 to 1.04]
Statistical Analysis 16: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 16]; Test type: Superiority or Other; p = 0.9872, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.00, 95% CI 2-sided [0.84 to 1.19]
Statistical Analysis 17: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 17]; Test type: Superiority or Other; p = 0.2582, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.85, 95% CI 2-sided [0.73 to 1.00]
Statistical Analysis 18: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 18]; Test type: Superiority or Other; p = 0.7918, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.06, 95% CI 2-sided [0.91 to 1.23]
Statistical Analysis 19: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 19]; Test type: Superiority or Other; p = 0.2514, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.86, 95% CI 2-sided [0.74 to 1.00]
Statistical Analysis 20: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 20]; Test type: Superiority or Other; p = 0.9765, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.03, 95% CI 2-sided [0.88 to 1.20]
Statistical Analysis 21: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 21]; Test type: Superiority or Other; p = 0.6915, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.06, 95% CI 2-sided [0.86 to 1.30]
Statistical Analysis 22: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 22]; Test type: Superiority or Other; p = 0.7918, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.13, 95% CI 2-sided [0.93 to 1.38]
Statistical Analysis 23: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 23]; Test type: Superiority or Other; p = 0.6922, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.95, 95% CI 2-sided [0.78 to 1.15]
Statistical Analysis 24: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 24]; Test type: Superiority or Other; p = 0.9872, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.01, 95% CI 2-sided [0.83 to 1.23]
Statistical Analysis 25: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 25]; Test type: Superiority or Other; p = 0.3609, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.85, 95% CI 2-sided [0.70 to 1.04]
Statistical Analysis 26: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 26]; Test type: Superiority or Other; p = 0.7918, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.08, 95% CI 2-sided [0.89 to 1.30]
Statistical Analysis 27: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 27]; Test type: Superiority or Other; p = 0.2514, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.86, 95% CI 2-sided [0.71 to 1.05]
Statistical Analysis 28: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 28]; Test type: Superiority or Other; p = 0.9765, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.04, 95% CI 2-sided [0.86 to 1.26]
Statistical Analysis 29: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 29]; Test type: Superiority or Other; p = 0.6304, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.92, 95% CI 2-sided [0.79 to 1.08]
Statistical Analysis 30: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 30]; Test type: Superiority or Other; p = 0.7918, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.06, 95% CI 2-sided [0.91 to 1.24]
Statistical Analysis 31: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 31]; Test type: Superiority or Other; p = 0.2514, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.88, 95% CI 2-sided [0.75 to 1.03]
Statistical Analysis 32: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 32]; Test type: Superiority or Other; p = 0.9765, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.03, 95% CI 2-sided [0.88 to 1.20]
Statistical Analysis 33: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 33]; Test type: Superiority or Other; p = 0.2582, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.84, 95% CI 2-sided [0.71 to 1.01]
Statistical Analysis 34: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 34]; Test type: Superiority or Other; p = 0.9279, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.99, 95% CI 2-sided [0.84 to 1.18]
Statistical Analysis 35: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 35]; Test type: Superiority or Other; p = 0.2514, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.85, 95% CI 2-sided [0.72 to 1.01]
Statistical Analysis 36: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 36]; Test type: Superiority or Other; p = 0.9765, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.90, 95% CI 2-sided [0.76 to 1.07]
Statistical Analysis 37: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 37]; Test type: Superiority or Other; p = 0.1424, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.82, 95% CI 2-sided [0.71 to 0.96]
Statistical Analysis 38: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 38]; Test type: Superiority or Other; p = 0.7918, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.97, 95% CI 2-sided [0.84 to 1.12]
Statistical Analysis 39: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 39]; Test type: Superiority or Other; p = 0.2514, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.85, 95% CI 2-sided [0.73 to 0.98]
Statistical Analysis 40: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 40]; Test type: Superiority or Other; p = 0.9765, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.92, 95% CI 2-sided [0.79 to 1.07]
Statistical Analysis 41: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 41]; Test type: Superiority or Other; p = 0.6304, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.93, 95% CI 2-sided [0.78 to 1.10]
Statistical Analysis 42: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 42]; Test type: Superiority or Other; p = 0.7918, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.04, 95% CI 2-sided [0.88 to 1.22]
Statistical Analysis 43: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 43]; Test type: Superiority or Other; p = 0.6922, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.95, 95% CI 2-sided [0.81 to 1.13]
Statistical Analysis 44: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 44]; Test type: Superiority or Other; p = 0.9765, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.97, 95% CI 2-sided [0.82 to 1.15]
Statistical Analysis 45: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 45]; Test type: Superiority or Other; p = 0.6572, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.95, 95% CI 2-sided [0.84 to 1.08]
Statistical Analysis 46: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 46]; Test type: Superiority or Other; p = 0.7918, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.98, 95% CI 2-sided [0.86 to 1.11]
Statistical Analysis 47: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 47]; Test type: Superiority or Other; p = 0.2514, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.89, 95% CI 2-sided [0.79 to 1.01]
Statistical Analysis 48: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 48]; Test type: Superiority or Other; p = 0.9872, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.00, 95% CI 2-sided [0.88 to 1.13]
Statistical Analysis 49: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 49]; Test type: Superiority or Other; p = 0.6304, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.92, 95% CI 2-sided [0.78 to 1.09]
Statistical Analysis 50: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 50]; Test type: Superiority or Other; p = 0.7918, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.04, 95% CI 2-sided [0.88 to 1.22]
Statistical Analysis 51: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 51]; Test type: Superiority or Other; p = 0.6922, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.95, 95% CI 2-sided [0.80 to 1.12]
Statistical Analysis 52: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 1, analysis 52]; Test type: Superiority or Other; p = 0.9765, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.95, 95% CI 2-sided [0.81 to 1.13]

4. Secondary Outcome: Percentage of Participants Achieving Serotype-Specific Pneumococcal Opsonophagocytic Activity (OPA) Titers Greater Than or Equal to (>=) Lower Limit of Quantitation (LLOQ) 1 Month After the Infant Series
Description: Percentage of participants achieving serotype-specific pneumococcal OPA titer >= LLOQ, along with the corresponding 95% CIs for 13 pneumococcal serotypes (4, 6B, 9V, 14, 18C, 19F, 23F, 1, 3, 5, 6A, 7F and 19A) are presented. Exact 2-sided CI based on the observed proportion of participants. The OPA LLOQ in titers for each serotype: 1 = 1:18; 3 = 1:12; 4 = 1:21; 5 = 1:29; 6A = 1:37; 6B = 1:43; 7F = 1:210; 9V = 1:345; 14 = 1:35; 18C = 1:31; 19A = 1:18; 19F = 1:48; 23F = 1:13.
Time Frame: 1 month after the infant series
Population: mITT infant immunogenicity population. Here 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure and 'n' signifies participants with a determinate IgG concentration to the given serotype for each arm respectively.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily | 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily | 13vPnC + INFANRIX Hexa
Number analyzed (Participants) | 46 | 48 | 44 | 44 | 76
percentage of participants
  4 (n = 37, 46, 42, 41, 61) | 100.0 [90.5 to 100.0] | 100.0 [92.3 to 100.0] | 100.0 [91.6 to 100.0] | 100.0 [91.4 to 100.0] | 100.0 [94.1 to 100.0]
  6B (n = 36, 45, 43, 40, 62) | 94.4 [81.3 to 99.3] | 88.9 [75.9 to 96.3] | 88.4 [74.9 to 96.1] | 92.5 [79.6 to 98.4] | 96.8 [88.8 to 99.6]
  9V (n = 37, 48, 42, 41, 65) | 62.2 [44.8 to 77.5] | 66.7 [51.6 to 79.6] | 59.5 [43.3 to 74.4] | 80.5 [65.1 to 91.2] | 75.4 [63.1 to 85.2]
  14 (n = 38, 48, 41, 41, 64) | 89.5 [75.2 to 97.1] | 97.9 [88.9 to 99.9] | 100.0 [91.4 to 100.0] | 97.6 [87.1 to 99.9] | 96.9 [89.2 to 99.6]
  18C (n = 37, 47, 41, 41, 62) | 100.0 [90.5 to 100.0] | 95.7 [85.5 to 99.5] | 100.0 [91.4 to 100.0] | 97.6 [87.1 to 99.9] | 100.0 [94.2 to 100.0]
  19F (n = 37, 46, 41, 42, 63) | 97.3 [85.8 to 99.9] | 87.0 [73.7 to 95.1] | 90.2 [76.9 to 97.3] | 92.9 [80.5 to 98.5] | 95.2 [86.7 to 99.0]
  23F (n = 38, 45, 42, 42, 63) | 92.1 [78.6 to 98.3] | 97.8 [88.2 to 99.9] | 92.9 [80.5 to 98.5] | 90.5 [77.4 to 97.3] | 93.7 [84.5 to 98.2]
  1 (n = 42, 42, 43, 44, 74) | 47.6 [32.0 to 63.6] | 42.9 [27.7 to 59.0] | 30.2 [17.2 to 46.1] | 29.5 [16.8 to 45.2] | 45.9 [34.3 to 57.9]
  3 (n = 41, 41, 39, 39, 69) | 97.6 [87.1 to 99.9] | 97.6 [87.1 to 99.9] | 97.4 [86.5 to 99.9] | 94.9 [82.7 to 99.4] | 100.0 [94.8 to 100.0]
  5 (n = 42, 43, 44, 42, 73) | 92.9 [80.5 to 98.5] | 90.7 [77.9 to 97.4] | 86.4 [72.6 to 94.8] | 92.9 [80.5 to 98.5] | 86.3 [76.2 to 93.2]
  6A (n = 46, 42, 39, 39, 76) | 93.5 [82.1 to 98.6] | 100.0 [91.6 to 100.0] | 100.0 [91.0 to 100.0] | 100.0 [91.0 to 100.0] | 98.7 [92.9 to 100.0]
  7F (n = 46, 42, 40, 39, 76) | 100.0 [92.3 to 100.0] | 100.0 [91.6 to 100.0] | 100.0 [91.2 to 100.0] | 97.4 [86.5 to 99.9] | 100.0 [95.3 to 100.0]
  19A (n = 42, 44, 41, 42, 74) | 92.9 [80.5 to 98.5] | 100.0 [92.0 to 100.0] | 90.2 [76.9 to 97.3] | 88.1 [74.4 to 96.0] | 97.3 [90.6 to 99.7]

5. Secondary Outcome: Geometric Mean Titer (GMT) for Serotype-specific Pneumococcal Opsonophagocytic Activity (OPA) 1 Month After the Infant Series
Description: Antibody-mediated serum OPA against the 13 pneumococcal serotypes (4, 6B, 9V, 14, 18C, 19F, 23F, 1, 3, 5, 6A, 7F and 19A) was measured centrally using a pneumococcal OPA assay. Results were expressed as OPA titers. OPA titers were logarithmically transformed for analysis; geometric means calculated and expressed as geometric mean titers (GMTs).
Time Frame: 1 month after the infant series
Population: mITT infant immunogenicity population. Here 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure and 'n' signifies participants with a determinate OPA titer to the given serotype for each arm respectively.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily | 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily | 13vPnC + INFANRIX Hexa
Number analyzed (Participants) | 46 | 48 | 44 | 44 | 76
titer
  4 (n = 37, 46, 42, 41, 61) | 1269 [961.2 to 1674.2] | 1135 [885.2 to 1456.1] | 1240 [955.9 to 1609.3] | 1361 [1045.4 to 1771.0] | 1086 [874.9 to 1347.9]
  6B (n = 36, 45, 43, 40, 62) | 794 [450.4 to 1399.6] | 655 [394.6 to 1087.9] | 470 [279.9 to 789.7] | 663 [387.2 to 1135.1] | 748 [485.6 to 1152.0]
  9V (n = 37, 48, 42, 41, 65) | 120 [52.5 to 274.2] | 166 [80.5 to 343.3] | 93 [43.0 to 203.0] | 285 [129.8 to 623.8] | 241 [129.0 to 448.7]
  14 (n = 38, 48, 41, 41, 64) | 435 [277.2 to 683.5] | 622 [416.0 to 928.6] | 650 [420.7 to 1003.0] | 991 [642.1 to 1530.9] | 951 [671.6 to 1346.3]
  18C (n = 37, 47, 41, 41, 62) | 1094 [777.8 to 1539.2] | 853 [630.0 to 1154.3] | 877 [634.1 to 1212.7] | 1031 [745.8 to 1426.2] | 1092 [838.9 to 1421.3]
  19F (n = 37, 46, 41, 42, 63) | 346 [219.7 to 545.4] | 221 [146.8 to 331.9] | 165 [106.8 to 253.4] | 294 [191.8 to 450.2] | 279 [196.8 to 395.0]
  23F (n = 38, 45, 42, 42, 63) | 342 [211.6 to 552.6] | 441 [283.7 to 685.4] | 332 [210.0 to 523.4] | 321 [203.3 to 506.7] | 366 [252.4 to 532.1]
  1 (n = 42, 42, 43, 44, 74) | 12 [8.7 to 17.7] | 11 [7.5 to 15.4] | 8 [5.5 to 11.2] | 8 [5.4 to 10.9] | 12 [9.0 to 15.5]
  3 (n = 41, 41, 39, 39, 69) | 72 [57.4 to 91.1] | 76 [60.4 to 95.7] | 56 [44.1 to 70.8] | 62 [49.3 to 79.1] | 87 [73.1 to 104.3]
  5 (n = 42, 43, 44, 42, 73) | 86 [59.7 to 122.7] | 96 [67.4 to 137.3] | 54 [37.7 to 76.2] | 99 [69.1 to 142.0] | 76 [57.5 to 99.2]
  6A (n = 46, 42, 39, 39, 76) | 1060 [784.5 to 1431.1] | 1681 [1227.3 to 2302.3] | 1228 [886.0 to 1701.9] | 1281 [924.0 to 1775.1] | 1462 [1157.1 to 1847.1]
  7F (n = 46, 42, 40, 39, 76) | 1766 [1387.0 to 2247.7] | 1907 [1481.0 to 2454.6] | 1747 [1348.6 to 2263.3] | 1584 [1218.8 to 2058.9] | 2125 [1761.6 to 2564.6]
  19A (n = 42, 44, 41, 42, 74) | 185 [127.8 to 268.3] | 257 [178.5 to 368.5] | 163 [112.3 to 237.9] | 159 [110.0 to 230.9] | 240 [181.9 to 318.0]
Statistical Analysis 1: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 4: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.7148, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 1.2, 95% CI 2-sided [0.82 to 1.66]
Statistical Analysis 2: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 4: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.7907, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 1.0, 95% CI 2-sided [0.75 to 1.45]
Statistical Analysis 3: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 4: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.4765, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 1.1, 95% CI 2-sided [0.81 to 1.60]
Statistical Analysis 4: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 4: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.5037, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 1.3, 95% CI 2-sided [0.89 to 1.76]
Statistical Analysis 5: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 6B: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.9414, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 1.1, 95% CI 2-sided [0.52 to 2.17]
Statistical Analysis 6: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 6B: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.7907, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.9, 95% CI 2-sided [0.45 to 1.71]
Statistical Analysis 7: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 6B: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.2900, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.6, 95% CI 2-sided [0.32 to 1.23]
Statistical Analysis 8: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 6B: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.8826, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.9, 95% CI 2-sided [0.44 to 1.77]
Statistical Analysis 9: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 9V: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.5823, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.5, 95% CI 2-sided [0.18 to 1.40]
Statistical Analysis 10: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 9V: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.7636, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.7, 95% CI 2-sided [0.27 to 1.80]
Statistical Analysis 11: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 9V: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.2407, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.4, 95% CI 2-sided [0.14 to 1.05]
Statistical Analysis 12: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 9V: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.8826, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 1.2, 95% CI 2-sided [0.43 to 3.22]
Statistical Analysis 13: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 14: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.0961, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.5, 95% CI 2-sided [0.26 to 0.81]
Statistical Analysis 14: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 14: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.7636, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.7, 95% CI 2-sided [0.38 to 1.11]
Statistical Analysis 15: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 14: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.2900, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.7, 95% CI 2-sided [0.39 to 1.19]
Statistical Analysis 16: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 14: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.8826, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 1.0, 95% CI 2-sided [0.60 to 1.82]
Statistical Analysis 17: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 18C: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.9925, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 1.0, 95% CI 2-sided [0.65 to 1.54]
Statistical Analysis 18: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 18C: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.7636, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.8, 95% CI 2-sided [0.52 to 1.17]
Statistical Analysis 19: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 18C: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.3929, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.8, 95% CI 2-sided [0.53 to 1.22]
Statistical Analysis 20: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 18C: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.8826, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.9, 95% CI 2-sided [0.62 to 1.43]
Statistical Analysis 21: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 19F: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.7433, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 1.2, 95% CI 2-sided [0.70 to 2.20]
Statistical Analysis 22: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 19F: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.7636, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.8, 95% CI 2-sided [0.46 to 1.35]
Statistical Analysis 23: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 19F: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.2407, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.6, 95% CI 2-sided [0.34 to 1.03]
Statistical Analysis 24: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 19F: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.8826, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 1.1, 95% CI 2-sided [0.61 to 1.83]
Statistical Analysis 25: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 23F: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.9414, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.9, 95% CI 2-sided [0.51 to 1.71]
Statistical Analysis 26: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 23F: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.7636, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 1.2, 95% CI 2-sided [0.68 to 2.14]
Statistical Analysis 27: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 23F: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.7380, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.9, 95% CI 2-sided [0.50 to 1.63]
Statistical Analysis 28: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 23F: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.8826, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.9, 95% CI 2-sided [0.49 to 1.58]
Statistical Analysis 29: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 1: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.9414, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 1.1, 95% CI 2-sided [0.67 to 1.65]
Statistical Analysis 30: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 1: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.7907, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.9, 95% CI 2-sided [0.58 to 1.43]
Statistical Analysis 31: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 1: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.2407, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.7, 95% CI 2-sided [0.43 to 1.04]
Statistical Analysis 32: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 1: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.2670, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.7, 95% CI 2-sided [0.42 to 1.02]
Statistical Analysis 33: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 3: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.5823, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.8, 95% CI 2-sided [0.62 to 1.11]
Statistical Analysis 34: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 3: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.7636, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.9, 95% CI 2-sided [0.65 to 1.16]
Statistical Analysis 35: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 3: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.0422, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.6, 95% CI 2-sided [0.48 to 0.86]
Statistical Analysis 36: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 3: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.2670, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.7, 95% CI 2-sided [0.53 to 0.96]
Statistical Analysis 37: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 5: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.8454, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 1.1, 95% CI 2-sided [0.72 to 1.78]
Statistical Analysis 38: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 5: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.7636, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 1.3, 95% CI 2-sided [0.81 to 2.00]
Statistical Analysis 39: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 5: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.2824, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.7, 95% CI 2-sided [0.45 to 1.11]
Statistical Analysis 40: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 5: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.5155, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 1.3, 95% CI 2-sided [0.83 to 2.06]
Statistical Analysis 41: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 6A: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.5823, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.7, 95% CI 2-sided [0.50 to 1.06]
Statistical Analysis 42: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 6A: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.7636, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 1.1, 95% CI 2-sided [0.78 to 1.70]
Statistical Analysis 43: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 6A: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.4644, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.8, 95% CI 2-sided [0.56 to 1.25]
Statistical Analysis 44: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 6A: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.8826, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.9, 95% CI 2-sided [0.59 to 1.31]
Statistical Analysis 45: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 7F: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.5823, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.8, 95% CI 2-sided [0.61 to 1.13]
Statistical Analysis 46: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 7F: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.7636, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.9, 95% CI 2-sided [0.65 to 1.23]
Statistical Analysis 47: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 7F: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.3299, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.8, 95% CI 2-sided [0.60 to 1.13]
Statistical Analysis 48: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 7F: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.2670, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.7, 95% CI 2-sided [0.54 to 1.03]
Statistical Analysis 49: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 19A: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.5823, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.8, 95% CI 2-sided [0.48 to 1.23]
Statistical Analysis 50: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; Serotype 19A: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.7907, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 1.1, 95% CI 2-sided [0.68 to 1.69]
Statistical Analysis 51: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 19A: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.2742, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.7, 95% CI 2-sided [0.43 to 1.09]
Statistical Analysis 52: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; Serotype 19A: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.2670, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.7, 95% CI 2-sided [0.42 to 1.05]

6. Secondary Outcome: Geometric Mean Concentration (GMC) for Antigen-specific Haemophilus Influenzae Type b (Hib) Polyribosylribitol Phosphate (PRP) Antibody 1 Month After the Infant Series
Description: Geometric LS mean concentrations (GMCs) and corresponding 2-sided 95% CIs were evaluated for Hib PRP antibody.
Time Frame: 1 month after the infant series
Population: mITT infant immunogenicity population. Here 'N' (number of participants analyzed) signifies participants with a determinate antibody concentration to the given concomitant vaccine antigen.
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily | 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily | 13vPnC + INFANRIX Hexa
Number analyzed (Participants) | 136 | 146 | 144 | 139 | 198
mcg/mL | 0.54 [0.44 to 0.66] | 0.59 [0.49 to 0.73] | 0.49 [0.40 to 0.60] | 0.51 [0.42 to 0.63] | 0.58 [0.49 to 0.69]
Statistical Analysis 1: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; Ratio of GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.813, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.93, 95% CI 2-sided [0.71 to 1.22]
Statistical Analysis 2: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; Ratio of GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.845, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.03, 95% CI 2-sided [0.79 to 1.34]
Statistical Analysis 3: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; Ratio of GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.461, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.85, 95% CI 2-sided [0.65 to 1.11]
Statistical Analysis 4: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; Ratio of GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.545, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.89, 95% CI 2-sided [0.68 to 1.16]

7. Secondary Outcome: Geometric Mean Concentration (GMC) for Antigen-specific Pertussis Toxin (PT), Filamentous Hemagglutinin (FHA) and Pertactin (PRN) Antibody 1 Month After the Infant Series
Description: Geometric LS mean concentration (GMCs) were measured in Enzyme-linked Immunosorbent Assay (ELISA) units/mL (EU/mL) and corresponding 2-sided 95% CIs were evaluated for pertussis (pertussis toxin [PT], filamentous hemagglutinin [FHA] and pertactin [PRN]) antibodies.
Time Frame: 1 month after the infant series
Population: mITT infant immunogenicity population. Here 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily | 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily | 13vPnC + INFANRIX Hexa
Number analyzed (Participants) | 132 | 143 | 141 | 131 | 193
EU/mL
  Pertussis PT | 40.86 [36.49 to 45.76] | 43.51 [39.02 to 48.51] | 40.27 [36.09 to 44.93] | 39.26 [35.04 to 43.98] | 44.85 [40.84 to 49.25]
  Pertussis FHA | 46.29 [41.49 to 51.65] | 40.65 [36.59 to 45.16] | 41.32 [37.16 to 45.94] | 35.55 [31.85 to 39.68] | 48.42 [44.22 to 53.01]
  Pertussis PRN | 72.90 [63.26 to 84.01] | 71.26 [62.18 to 81.66] | 65.82 [57.38 to 75.50] | 68.53 [59.44 to 79.02] | 84.57 [75.21 to 95.09]
Statistical Analysis 1: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; Pertussis PT: Ratio of GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.712, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.91, 95% CI 2-sided [0.79 to 1.06]
Statistical Analysis 2: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; Pertussis PT: Ratio of GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.837, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.97, 95% CI 2-sided [0.84 to 1.12]
Statistical Analysis 3: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; Pertussis PT: Ratio of GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.357, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.90, 95% CI 2-sided [0.78 to 1.04]
Statistical Analysis 4: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; Pertussis PT: Ratio of GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.190, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.88, 95% CI 2-sided [0.76 to 1.01]
Statistical Analysis 5: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; Pertussis FHA: Ratio of GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.813, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.96, 95% CI 2-sided [0.83 to 1.10]
Statistical Analysis 6: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; Pertussis FHA: Ratio of GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.136, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.84, 95% CI 2-sided [0.73 to 0.96]
Statistical Analysis 7: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; Pertussis FHA: Ratio of GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.104, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.85, 95% CI 2-sided [0.74 to 0.98]
Statistical Analysis 8: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; Pertussis FHA: Ratio of GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p < 0.001, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.73, 95% CI 2-sided [0.64 to 0.85]
Statistical Analysis 9: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; Pertussis PRN: Ratio of GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.712, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.86, 95% CI 2-sided [0.72 to 1.04]
Statistical Analysis 10: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; Pertussis PRN: Ratio of GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.206, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.84, 95% CI 2-sided [0.70 to 1.01]
Statistical Analysis 11: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; Pertussis PRN: Ratio of GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.066, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.78, 95% CI 2-sided [0.65 to 0.93]
Statistical Analysis 12: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; Pertussis PRN: Ratio of GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.085, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.81, 95% CI 2-sided [0.67 to 0.97]

8. Secondary Outcome: Geometric Mean Concentration (GMC) for Antigen-specific Tetanus and Diphtheria Antibody 1 Month After the Infant Series
Description: Geometric LS mean concentration (GMCs) were measured in International Units/mL (IU/mL) and corresponding 2-sided 95% CIs were evaluated for tetanus and diphtheria antibodies.
Time Frame: 1 month after the infant series
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily | 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily | 13vPnC + INFANRIX Hexa
Number analyzed (Participants) | 132 | 143 | 141 | 131 | 193
IU/mL
  Tetanus | 0.73 [0.65 to 0.83] | 0.70 [0.62 to 0.79] | 0.69 [0.61 to 0.77] | 0.60 [0.53 to 0.68] | 0.82 [0.74 to 0.90]
  Diphtheria | 0.62 [0.56 to 0.69] | 0.68 [0.61 to 0.75] | 0.61 [0.55 to 0.68] | 0.65 [0.59 to 0.73] | 0.65 [0.60 to 0.72]
Statistical Analysis 1: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; Tetanus: Ratio of GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.712, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.90, 95% CI 2-sided [0.77 to 1.06]
Statistical Analysis 2: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; Tetanus: Ratio of GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.206, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.86, 95% CI 2-sided [0.74 to 1.00]
Statistical Analysis 3: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; Tetanus: Ratio of GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.104, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.84, 95% CI 2-sided [0.72 to 0.98]
Statistical Analysis 4: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; Tetanus: Ratio of GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.001, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.74, 95% CI 2-sided [0.63 to 0.87]
Statistical Analysis 5: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; Diphtheria: Ratio of GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.813, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.95, 95% CI 2-sided [0.82 to 1.09]
Statistical Analysis 6: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; Diphtheria: Ratio of GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.837, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.03, 95% CI 2-sided [0.90 to 1.19]
Statistical Analysis 7: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; Diphtheria: Ratio of GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.534, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.93, 95% CI 2-sided [0.81 to 1.07]
Statistical Analysis 8: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; Diphtheria: Ratio of GMCs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.961, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.00, 95% CI 2-sided [0.87 to 1.15]

9. Secondary Outcome: Geometric Mean Concentration (GMC) for Antigen-specific Hepatitis B Virus (HBV) Antibody 1 Month After the Infant Series
Description: Geometric LS mean concentration (GMCs) were measured in milli international units/mL (mIU/mL) and corresponding 2-sided 95% CIs were evaluated for hepatitis B virus (HBV) antibody.
Time Frame: 1 month after the infant series
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily | 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily | 13vPnC + INFANRIX Hexa
Number analyzed (Participants) | 105 | 116 | 120 | 112 | 156
mIU/mL | 756.42 [589.71 to 970.26] | 770.93 [608.34 to 976.98] | 689.34 [546.12 to 870.11] | 599.12 [470.78 to 762.43] | 733.29 [597.81 to 899.46]
Statistical Analysis 1: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.850, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.03, 95% CI 2-sided [0.75 to 1.42]
Statistical Analysis 2: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 6, analysis 2]; Test type: Superiority or Other; p = 0.837, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.05, 95% CI 2-sided [0.77 to 1.44]
Statistical Analysis 3: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 6, analysis 3]; Test type: Superiority or Other; p = 0.695, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.94, 95% CI 2-sided [0.69 to 1.28]
Statistical Analysis 4: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p = 0.408, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.82, 95% CI 2-sided [0.60 to 1.12]

10. Secondary Outcome: Geometric Mean Titer (GMT) for Antigen-specific Poliomyelitis Type 1, 2 and 3 Antibodies 1 Month After the Infant Series
Description: Geometric LS mean concentrations (GMCs) were measured as titers and corresponding 2-sided 95% CIs were evaluated for poliomyelitis type 1, 2 and 3 antibodies.
Time Frame: 1 month after the infant series
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily | 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily | 13vPnC + INFANRIX Hexa
Number analyzed (Participants) | 89 | 105 | 93 | 84 | 135
titer
  Poliomyelitis Type 1 | 68.11 [53.14 to 87.30] | 66.59 [52.98 to 83.68] | 67.43 [52.89 to 85.96] | 70.66 [54.73 to 91.23] | 72.02 [58.88 to 88.10]
  Poliomyelitis Type 2 | 79.60 [61.54 to 102.95] | 73.52 [58.01 to 93.16] | 62.12 [48.30 to 79.90] | 55.17 [42.33 to 71.89] | 67.37 [54.67 to 83.02]
  Poliomyelitis Type 3 | 246.22 [192.84 to 314.38] | 184.03 [146.96 to 230.46] | 257.92 [203.08 to 327.56] | 218.85 [170.18 to 281.44] | 231.02 [189.44 to 281.72]
Statistical Analysis 1: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; Poliomyelitis Type 1: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.813, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.95, 95% CI 2-sided [0.69 to 1.30]
Statistical Analysis 2: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; Poliomyelitis Type 1: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.837, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.92, 95% CI 2-sided [0.68 to 1.25]
Statistical Analysis 3: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; Poliomyelitis Type 1: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.695, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.94, 95% CI 2-sided [0.68 to 1.28]
Statistical Analysis 4: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; Poliomyelitis Type 1: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.961, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.98, 95% CI 2-sided [0.71 to 1.36]
Statistical Analysis 5: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; Poliomyelitis Type 2: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.808, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 1.18, 95% CI 2-sided [0.85 to 1.65]
Statistical Analysis 6: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; Poliomyelitis Type 2: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.837, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 1.09, 95% CI 2-sided [0.80 to 1.50]
Statistical Analysis 7: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; Poliomyelitis Type 2: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.695, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.92, 95% CI 2-sided [0.66 to 1.28]
Statistical Analysis 8: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; Poliomyelitis Type 2: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.408, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.82, 95% CI 2-sided [0.58 to 1.15]
Statistical Analysis 9: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; Poliomyelitis Type 3: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.813, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 1.07, 95% CI 2-sided [0.78 to 1.46]
Statistical Analysis 10: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; Poliomyelitis Type 3: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen twice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.343, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.80, 95% CI 2-sided [0.59 to 1.08]
Statistical Analysis 11: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; Poliomyelitis Type 3: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Paracetamol thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.695, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 1.12, 95% CI 2-sided [0.82 to 1.52]
Statistical Analysis 12: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; Poliomyelitis Type 3: Ratio of GMTs along with 2-sided 95% CI were back transformed from the difference of the LS mean of 13vPnC + INFANRIX hexa + Ibuprofen thrice daily group minus the LS mean of 13vPnC + INFANRIX hexa group; Test type: Superiority or Other; p = 0.925, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.95, 95% CI 2-sided [0.69 to 1.31]

11. Secondary Outcome: Geometric Mean Concentration (GMC) for Antigen-specific Haemophilus Influenzae Type b (Hib) Polyribosylribitol Phosphate (PRP) Antibody 1 Month After the Toddler Dose
Description: Geometric LS mean concentration (GMCs) were measured in mcg/mL and corresponding 2-sided 95% CIs were evaluated for Hib PRP antibody.
Time Frame: 1 month after the toddler dose
Population: mITT toddler immunogenicity population. Here 'N' (number of participants analyzed) signifies participants with a determinate antibody concentration to the given concomitant vaccine antigen.
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily | 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily | 13vPnC + INFANRIX Hexa
Number analyzed (Participants) | 126 | 135 | 141 | 138 | 202
mcg/mL | 9.65 [7.74 to 12.03] | 9.35 [7.55 to 11.57] | 8.25 [6.69 to 10.16] | 7.84 [6.35 to 9.68] | 8.96 [7.53 to 10.67]
Statistical Analysis 1: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.910, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.08, 95% CI 2-sided [0.81 to 1.43]
Statistical Analysis 2: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 6, analysis 2]; Test type: Superiority or Other; p = 0.850, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.04, 95% CI 2-sided [0.79 to 1.37]
Statistical Analysis 3: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 6, analysis 3]; Test type: Superiority or Other; p = 0.868, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.92, 95% CI 2-sided [0.70 to 1.21]
Statistical Analysis 4: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p = 0.914, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.87, 95% CI 2-sided [0.67 to 1.15]

12. Secondary Outcome: Geometric Mean Concentration (GMC) for Antigen-specific Pertussis Toxin (PT), Filamentous Hemagglutinin (FHA) and Pertactin (PRN) Antibodies 1 Month After the Toddler Dose
Description: Geometric LS mean concentration (GMCs) were measured in EU/mL and corresponding 2-sided 95% CIs were evaluated for pertussis (pertussis toxin [PT], filamentous hemagglutinin [FHA] and pertactin [PRN]) antibodies.
Time Frame: 1 month after the toddler dose
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily | 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily | 13vPnC + INFANRIX Hexa
Number analyzed (Participants) | 123 | 137 | 141 | 136 | 199
EU/mL
  Pertussis PT | 77.43 [68.12 to 88.02] | 76.93 [68.13 to 86.87] | 73.72 [65.40 to 83.10] | 73.38 [64.96 to 82.90] | 74.01 [66.91 to 81.86]
  Pertussis FHA | 115.55 [104.32 to 128.00] | 117.87 [106.98 to 129.87] | 123.56 [112.30 to 135.95] | 108.11 [98.09 to 119.16] | 117.01 [107.97 to 126.81]
  Pertussis PRN | 158.28 [136.30 to 183.81] | 156.98 [136.24 to 180.87] | 160.96 [139.98 to 185.08] | 158.71 [137.67 to 182.97] | 172.80 [153.64 to 194.36]
Statistical Analysis 1: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.910, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.05, 95% CI 2-sided [0.89 to 1.23]
Statistical Analysis 2: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; p = 0.850, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.04, 95% CI 2-sided [0.89 to 1.22]
Statistical Analysis 3: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 7, analysis 3]; Test type: Superiority or Other; p = 0.961, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.00, 95% CI 2-sided [0.85 to 1.16]
Statistical Analysis 4: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 7, analysis 4]; Test type: Superiority or Other; p = 0.916, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.99, 95% CI 2-sided [0.85 to 1.16]
Statistical Analysis 5: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 7, analysis 5]; Test type: Superiority or Other; p = 0.910, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.99, 95% CI 2-sided [0.87 to 1.12]
Statistical Analysis 6: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 7, analysis 6]; Test type: Superiority or Other; p = 0.909, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.01, 95% CI 2-sided [0.89 to 1.14]
Statistical Analysis 7: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; p = 0.868, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.06, 95% CI 2-sided [0.93 to 1.20]
Statistical Analysis 8: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 7, analysis 8]; Test type: Superiority or Other; p = 0.914, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.92, 95% CI 2-sided [0.81 to 1.05]
Statistical Analysis 9: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 7, analysis 9]; Test type: Superiority or Other; p = 0.910, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.92, 95% CI 2-sided [0.76 to 1.11]
Statistical Analysis 10: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 7, analysis 10]; Test type: Superiority or Other; p = 0.850, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.91, 95% CI 2-sided [0.76 to 1.09]
Statistical Analysis 11: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 7, analysis 11]; Test type: Superiority or Other; p = 0.868, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.93, 95% CI 2-sided [0.78 to 1.12]
Statistical Analysis 12: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 7, analysis 12]; Test type: Superiority or Other; p = 0.914, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.92, 95% CI 2-sided [0.76 to 1.10]

13. Secondary Outcome: Geometric Mean Concentration (GMC) for Antigen-specific Tetanus and Diphtheria Antibodies 1 Month After the Toddler Dose
Description: Geometric LS mean concentration (GMCs) were measured in IU/mL and corresponding 2-sided 95% CIs were evaluated for tetanus and diphtheria antibodies.
Time Frame: 1 month after the toddler dose
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily | 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily | 13vPnC + INFANRIX Hexa
Number analyzed (Participants) | 123 | 137 | 141 | 136 | 199
IU/mL
  Tetanus | 2.54 [2.28 to 2.83] | 2.50 [2.26 to 2.77] | 2.60 [2.35 to 2.88] | 2.29 [2.07 to 2.54] | 2.66 [2.44 to 2.89]
  Diphtheria | 1.64 [1.49 to 1.80] | 1.94 [1.77 to 2.12] | 1.69 [1.54 to 1.84] | 1.87 [1.71 to 2.04] | 1.90 [1.77 to 2.05]
Statistical Analysis 1: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.910, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.96, 95% CI 2-sided [0.83 to 1.10]
Statistical Analysis 2: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 8, analysis 2]; Test type: Superiority or Other; p = 0.850, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.94, 95% CI 2-sided [0.82 to 1.07]
Statistical Analysis 3: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 8, analysis 3]; Test type: Superiority or Other; p = 0.939, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.98, 95% CI 2-sided [0.86 to 1.12]
Statistical Analysis 4: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 8, analysis 4]; Test type: Superiority or Other; p = 0.279, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.86, 95% CI 2-sided [0.75 to 0.98]
Statistical Analysis 5: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 8, analysis 5]; Test type: Superiority or Other; p = 0.149, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.86, 95% CI 2-sided [0.76 to 0.97]
Statistical Analysis 6: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 8, analysis 6]; Test type: Superiority or Other; p = 0.850, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.02, 95% CI 2-sided [0.91 to 1.14]
Statistical Analysis 7: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 8, analysis 7]; Test type: Superiority or Other; p = 0.394, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.89, 95% CI 2-sided [0.79 to 0.99]
Statistical Analysis 8: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 8, analysis 8]; Test type: Superiority or Other; p = 0.916, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 0.98, 95% CI 2-sided [0.87 to 1.10]

14. Secondary Outcome: Geometric Mean Concentration (GMC) for Antigen-specific Hepatitis B Virus (HBV) Antibody 1 Month After the Toddler Dose
Description: Geometric LS mean concentration (GMCs) were measured in mIU/mL and corresponding 2-sided 95% CIs were evaluated for hepatitis B virus (HBV) antibody.
Time Frame: 1 month after the toddler dose
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily | 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily | 13vPnC + INFANRIX Hexa
Number analyzed (Participants) | 119 | 131 | 133 | 133 | 191
mIU/mL | 4868.61 [3750.57 to 6319.94] | 4148.04 [3234.82 to 5319.08] | 4250.41 [3320.88 to 5440.13] | 4263.28 [3330.93 to 5456.60] | 3866.37 [3146.78 to 4750.52]
Statistical Analysis 1: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.869, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.26, 95% CI 2-sided [0.90 to 1.76]
Statistical Analysis 2: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 6, analysis 2]; Test type: Superiority or Other; p = 0.850, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.07, 95% CI 2-sided [0.78 to 1.48]
Statistical Analysis 3: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 6, analysis 3]; Test type: Superiority or Other; p = 0.868, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.10, 95% CI 2-sided [0.80 to 1.52]
Statistical Analysis 4: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p = 0.916, General Linear Model — P-values were adjusted using false discovery rate procedure; GMC Ratio = 1.10, 95% CI 2-sided [0.80 to 1.52]

15. Secondary Outcome: Geometric Mean Titer (GMT) for Antigen-specific Poliomyelitis Type 1, 2 and 3 Antibodies 1 Month After the Toddler Dose
Description: Geometric LS mean concentration (GMCs) were measured as titers and corresponding 2-sided 95% CIs were evaluated for poliomyelitis type 1, 2 and 3 antibodies.
Time Frame: 1 month after the toddler dose
Population: mITT toddler immunogenicity population. Here 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily | 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily | 13vPnC + INFANRIX Hexa
Number analyzed (Participants) | 123 | 133 | 141 | 136 | 201
titer
  Poliomyelitis Type 1 | 399.56 [332.13 to 480.68] | 426.63 [357.15 to 509.62] | 443.97 [373.58 to 527.63] | 415.45 [348.48 to 495.29] | 406.37 [351.67 to 469.59]
  Poliomyelitis Type 2 | 613.18 [515.30 to 729.65] | 586.30 [496.01 to 693.03] | 587.56 [499.47 to 691.18] | 605.78 [513.44 to 714.73] | 621.07 [542.07 to 711.57]
  Poliomyelitis Type 3 | 1205.80 [1001.18 to 1452.24] | 1045.57 [874.35 to 1250.32] | 1210.29 [1017.32 to 1439.87] | 1187.11 [994.68 to 1416.76] | 1237.86 [1070.27 to 1431.70]
Statistical Analysis 1: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.910, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.98, 95% CI 2-sided [0.78 to 1.24]
Statistical Analysis 2: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 10, analysis 2]; Test type: Superiority or Other; p = 0.850, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 1.05, 95% CI 2-sided [0.83 to 1.32]
Statistical Analysis 3: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 10, analysis 3]; Test type: Superiority or Other; p = 0.868, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 1.09, 95% CI 2-sided [0.87 to 1.37]
Statistical Analysis 4: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 10, analysis 4]; Test type: Superiority or Other; p = 0.916, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 1.02, 95% CI 2-sided [0.81 to 1.28]
Statistical Analysis 5: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 10, analysis 5]; Test type: Superiority or Other; p = 0.910, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.99, 95% CI 2-sided [0.79 to 1.23]
Statistical Analysis 6: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 10, analysis 6]; Test type: Superiority or Other; p = 0.850, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.94, 95% CI 2-sided [0.76 to 1.17]
Statistical Analysis 7: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 10, analysis 7]; Test type: Superiority or Other; p = 0.868, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.95, 95% CI 2-sided [0.77 to 1.17]
Statistical Analysis 8: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 10, analysis 8]; Test type: Superiority or Other; p = 0.916, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.98, 95% CI 2-sided [0.79 to 1.21]
Statistical Analysis 9: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 10, analysis 9]; Test type: Superiority or Other; p = 0.910, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.97, 95% CI 2-sided [0.77 to 1.23]
Statistical Analysis 10: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 10, analysis 10]; Test type: Superiority or Other; p = 0.850, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.84, 95% CI 2-sided [0.67 to 1.06]
Statistical Analysis 11: Comparison: 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 10, analysis 11]; Test type: Superiority or Other; p = 0.939, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.98, 95% CI 2-sided [0.78 to 1.23]
Statistical Analysis 12: Comparison: 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily vs 13vPnC + INFANRIX Hexa; [analysis description as in outcome 10, analysis 12]; Test type: Superiority or Other; p = 0.916, General Linear Model — P-values were adjusted using false discovery rate procedure; GMT Ratio = 0.96, 95% CI 2-sided [0.76 to 1.21]

16. Secondary Outcome: Percentage of Participants Achieving Pre-specified Criteria for the Concomitant Antigens Contained in INFANRIX Hexa 1 Month After the Infant Series
Description: Percentage of participants achieving pre-specified criteria for concomitant antigens contained in INFANRIX hexa (Hib polyribosylribitol phosphate [PRP] >=0.15 mcg/mL; Hib PRP >=1 mcg/mL; Pertussis PT >=14.6 EU/mL, FHA >=16.1 EU/mL, PRN >=24.0 EU/mL; Tetanus >=0.1 IU/mL; Diphtheria >=0.1 IU/mL; HBV >=10 mIU/mL; Poliomyelitis Type 1, 2, 3 >=1:8 titer) along with the corresponding 95% CIs were presented. Exact 2-sided CI based on the observed proportion of participants. Pre-specified criteria for pertussis was the level that 95% of the participants achieved in 13vPnC + INFANRIX hexa group.
Time Frame: 1 month after the infant series
Population: mITT infant immunogenicity population. Here 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure and 'n' signifies participants with a determinate antibody concentration or titer to the given concomitant vaccine antigen for each arm respectively.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily | 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily | 13vPnC + INFANRIX Hexa
Number analyzed (Participants) | 136 | 146 | 144 | 139 | 198
percentage of participants
  Hib PRP >=0.15 mcg/mL (n= 136, 146, 144, 139, 198) | 87.5 [80.7 to 92.5] | 84.2 [77.3 to 89.7] | 86.1 [79.4 to 91.3] | 85.6 [78.7 to 91.0] | 87.9 [82.5 to 92.1]
  Hib PRP >=1 mcg/mL (n = 136, 146, 144, 139, 198) | 33.8 [25.9 to 42.4] | 37.0 [29.2 to 45.4] | 27.1 [20.0 to 35.1] | 28.1 [20.8 to 36.3] | 33.8 [27.3 to 40.9]
  Pertussis PT >=14.6 EU/mL (n= 132,143,141,131,193) | 93.2 [87.5 to 96.8] | 97.2 [93.0 to 99.2] | 91.5 [85.6 to 95.5] | 90.8 [84.5 to 95.2] | 95.3 [91.3 to 97.8]
  Pertussis FHA >=16.1 EU/mL (n=132,143,141,131,193) | 96.2 [91.4 to 98.8] | 92.3 [86.7 to 96.1] | 93.6 [88.2 to 97.0] | 88.5 [81.8 to 93.4] | 95.3 [91.3 to 97.8]
  Pertussis PRN >=24.0 EU/mL (n=132,143,141,131,193) | 90.9 [84.7 to 95.2] | 87.4 [80.8 to 92.4] | 88.7 [82.2 to 93.4] | 89.3 [82.7 to 94.0] | 95.3 [91.3 to 97.8]
  Tetanus >=0.1 IU/mL (n = 132,143,141,131,193) | 100.0 [97.2 to 100.00] | 100.0 [97.5 to 100.00] | 100.0 [97.4 to 100.00] | 98.5 [94.6 to 99.8] | 99.5 [97.1 to 100.0]
  Diphtheria >=0.1 IU/mL (n = 132,143,141,131,193) | 100.0 [97.2 to 100.00] | 98.6 [95.0 to 99.8] | 99.3 [96.1 to 100.0] | 97.7 [93.5 to 99.5] | 99.5 [97.1 to 100.0]
  HBV >= 10mIU/mL (n = 105,116,120,112,156) | 100.0 [96.5 to 100.0] | 99.1 [95.3 to 100.0] | 99.2 [95.4 to 100.0] | 99.1 [95.1 to 100.0] | 98.7 [95.4 to 99.8]
  PoliomyelitisType1 >=1:8titer (n=89,105,93,84,135) | 97.8 [92.1 to 99.7] | 98.1 [93.3 to 99.8] | 97.8 [92.4 to 99.7] | 100.0 [95.7 to 100.0] | 99.3 [95.9 to 100.0]
  PoliomyelitisType2 >=1:8titer (n=89,105,93,84,135) | 95.5 [88.9 to 98.8] | 98.1 [93.3 to 99.8] | 95.7 [89.4 to 98.8] | 96.4 [89.9 to 99.3] | 95.6 [90.6 to 98.4]
  PoliomyelitisType3 >=1:8titer (n=89,105,93,84,135) | 100.0 [95.9 to 100.0] | 100.0 [96.5 to 100.0] | 98.9 [94.2 to 100.0] | 98.8 [93.5 to 100.0] | 99.3 [95.9 to 100.0]

17. Secondary Outcome: Percentage of Participants Achieving Pre-specified Criteria for the Concomitant Antigens Contained in INFANRIX Hexa 1 Month After the Toddler Dose
Description: Percentage of participants achieving pre-specified criteria for concomitant antigens contained in INFANRIX hexa (Hib polyribosylribitol phosphate [PRP] >=0.15 mcg/mL; Hib PRP >=1 mcg/mL; Pertussis PT >=14.8 EU/mL, FHA >=46.5 EU/mL, PRN >=43.5 EU/mL; Tetanus >=0.1 IU/mL; Diphtheria >=0.1 IU/mL; HBV >=10 mIU/mL; Poliomyelitis Type 1, 2, 3 >=1:8 titer) along with the corresponding 95% CIs were presented. Exact 2-sided CI based on the observed proportion of participants. Pre-specified criteria for pertussis was the level that 95% of the participants achieved in 13vPnC + INFANRIX hexa group.
Time Frame: 1 month after the toddler dose
Population: mITT toddler immunogenicity population. Here 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure and 'n' signifies participants with a determinate antibody concentration or titer to the given concomitant vaccine antigen for each arm respectively.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily | 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily | 13vPnC + INFANRIX Hexa
Number analyzed (Participants) | 126 | 137 | 141 | 138 | 202
percentage of participants
  Hib PRP >=0.15 mcg/mL (n= 126, 135, 141, 138, 202) | 100.0 [97.1 to 100.0] | 99.3 [95.9 to 100.0] | 100.0 [97.4 to 100.0] | 100.0 [97.4 to 100.0] | 100.0 [98.2 to 100.0]
  Hib PRP >=1 mcg/mL (n = 126, 135, 141, 138, 202) | 95.2 [89.9 to 98.2] | 96.3 [91.6 to 98.8] | 95.7 [91.0 to 98.4] | 95.7 [90.8 to 98.4] | 95.0 [91.1 to 97.6]
  Pertussis PT >=14.8 EU/mL (n= 123,137,141,136,199) | 97.6 [93.0 to 99.5] | 99.3 [96.0 to 100.0] | 98.6 [95.0 to 99.8] | 100.0 [97.3 to 100.0] | 95.5 [91.6 to 97.9]
  Pertussis FHA >=46.5 EU/mL (n=123,137,141,136,199) | 91.1 [84.6 to 95.5] | 94.9 [89.8 to 97.9] | 93.6 [88.2 to 97.0] | 92.6 [86.9 to 96.4] | 95.5 [91.6 to 97.9]
  Pertussis PRN >=43.5 EU/mL (n=123,137,141,136,199) | 91.9 [85.6 to 96.0] | 94.9 [89.8 to 97.9] | 94.3 [89.1 to 97.5] | 94.1 [88.7 to 97.4] | 95.5 [91.6 to 97.9]
  Tetanus >=0.1 IU/mL (n = 123,137,141,136,199) | 100.0 [97.0 to 100.0] | 100.0 [97.3 to 100.0] | 100.0 [97.4 to 100.0] | 100.0 [97.3 to 100.0] | 100.0 [98.2 to 100.0]
  Diphtheria >=0.1 IU/mL (n = 123,137,141,136,199) | 100.0 [97.0 to 100.0] | 100.0 [97.3 to 100.0] | 100.0 [97.4 to 100.0] | 100.0 [97.3 to 100.0] | 100.0 [98.2 to 100.0]
  HBV >= 10 mIU/mL (n = 119,131,133,133,191) | 100.0 [96.9 to 100.0] | 98.5 [94.6 to 99.8] | 100.0 [97.3 to 100.0] | 100.0 [97.3 to 100.0] | 99.5 [97.1 to 100.0]
  Poliomyelitis 1 >=1:8titer (n=123,133,141,136,201) | 99.2 [95.6 to 100.0] | 100.0 [97.3 to 100.0] | 100.0 [97.4 to 100.0] | 100.0 [97.3 to 100.0] | 99.5 [97.3 to 100.0]
  Poliomyelitis 2 >=1:8titer (n=123,133,141,136,201) | 100.0 [97.0 to 100.0] | 100.0 [97.3 to 100.0] | 100.0 [97.4 to 100.0] | 100.0 [97.3 to 100.0] | 100.0 [98.2 to 100.0]
  Poliomyelitis 3 >=1:8titer (n=123,133,141,136,201) | 100.0 [97.0 to 100.0] | 100.0 [97.3 to 100.0] | 100.0 [97.4 to 100.0] | 100.0 [97.3 to 100.0] | 100.0 [98.2 to 100.0]

18. Secondary Outcome: Percentage of Participants Reporting Fever Within 4 Days: Infant Series Dose 1
Description: Participants' core (rectal) temperature was collected for 4 days after each vaccination using an electronic diary. Participants' temperature was collected at 6 to 8 hours after vaccination, 6 to 8 hours following that and coincidentally with antipyretic administration for groups receiving antipyretics. Temperature was recorded at bedtime daily for 3 following days (Day 2 to Day 4) and at any time during the 3 days when fever was suspected. The highest temperature for each day was recorded in the e-diary. Incidences of fever were presented in following categories: >=38 but <=39 degree Celsius (degree C), greater than (>) 39 but <=40 degree C and >40 degree C.
Time Frame: Within 4 days after infant series Dose 1
Population: Safety analysis set Dose 1: participants who received Dose 1 of 13vPnC/INFANRIX hexa in infant series, had Adverse Event (AE) or temperature data. 'N'(number of participants analyzed)=participants reported yes for >=1 day or no for all days, 'n'=participants reporting yes for >=1 day or no for all days for specified event for each arm respectively.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily | 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily | 13vPnC + INFANRIX Hexa
Number analyzed (Participants) | 149 | 157 | 147 | 155 | 187
percentage of participants
  Fever >=38, <=39 degree C (n= 149,157,147,155,187) | 32.9 | 45.2 | 18.4 | 34.2 | 41.7
  Fever >39, <=40 degree C (n = 138,145,137,146,170) | 1.4 | 1.4 | 0.7 | 0.7 | 1.2
  Fever >40 degree C (n = 138,145,137,146,170) | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

19. Secondary Outcome: Percentage of Participants Reporting Fever Within 4 Days: Infant Series Dose 2
Description: Participants' rectal temperature was collected for 4 days after each vaccination using an electronic diary. Participants' temperature was collected at 6 to 8 hours after vaccination, 6 to 8 hours following that and coincidentally with antipyretic administration for groups receiving antipyretics. Temperature was recorded at bedtime daily for 3 following days (Day 2 to Day 4) and at any time during the 3 days when fever was suspected. The highest temperature for each day was recorded in the e-diary. Incidences of fever were presented in following categories: >=38 but <=39 degree C, >39 but <=40 degree C and >40 degree C.
Time Frame: Within 4 days after infant series Dose 2
Population: Safety analysis set Dose 2: participants who received Dose 2 of 13vPnC/INFANRIX hexa in infant series and had AE or temperature data available. 'N' (number of participants analyzed) =participants reported yes for >=1 day or no for all days, 'n'=participants reporting yes for >=1 day or no for all days for specified event for each arm respectively.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily | 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily | 13vPnC + INFANRIX Hexa
Number analyzed (Participants) | 141 | 152 | 140 | 159 | 181
percentage of participants
  Fever >=38, <=39 degree C (n= 141,152,140,159,181) | 26.2 | 42.8 | 21.4 | 44.0 | 39.8
  Fever >39, <=40 degree C (n = 133,140,134,145,164) | 1.5 | 0.7 | 1.5 | 1.4 | 3.7
  Fever >40 degree C (n = 131,140,133,144,164) | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

20. Secondary Outcome: Percentage of Participants Reporting Fever Within 4 Days: Infant Series Dose 3
Description: Participants' rectal temperature was collected for 4 days after each vaccination using an electronic diary. Participants' temperature was collected at 6 to 8 hours after vaccination, 6 to 8 hours following that and coincidentally with antipyretic administration for groups receiving antipyretics. Temperature was recorded at bedtime daily for 3 following days (Day 2 to Day 4) and at any time during the 3 days when fever was suspected. The highest temperature for each day was recorded in the e-diary. Incidences of fever were presented in following categories: >=38 but <=39 degree C, >39 but <=40 degree C and >40 degree C. Report of fever >40 degrees C after 13vPnC Infant Series Dose 3 was confirmed as data entry error.
Time Frame: Within 4 days after infant series Dose 3
Population: Safety analysis set Dose 3: participants who received Dose 3 of 13vPnC/INFANRIX hexa in infant series and had AE or temperature data available. 'N' (number of participants analyzed) =participants reported yes for >=1 day or no for all days, 'n'=participants reporting yes for >=1 day or no for all days for specified event for each arm respectively.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily | 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily | 13vPnC + INFANRIX Hexa
Number analyzed (Participants) | 136 | 146 | 135 | 141 | 175
percentage of participants
  Fever >=38, <=39 degree C (n= 136,146,135,141,175) | 22.1 | 30.8 | 17.0 | 33.3 | 29.7
  Fever >39, <=40 degree C (n = 129,137,125,136,167) | 1.6 | 2.9 | 0.8 | 1.5 | 1.8
  Fever >40 degree C (n = 128,136,126,135,166) | 0.0 | 0.0 | 0.8 | 0.0 | 0.0

21. Secondary Outcome: Percentage of Participants Reporting Fever Within 4 Days: Toddler Dose
Description: as for outcome 19
Time Frame: Within 4 days after toddler dose
Population: Safety analysis set toddler dose: participants who receive toddler dose of 13vPnC or INFANRIX hexa and had AE or temperature data available. 'N' (number of participants analyzed) =participants reported yes for >=1 day or no for all days, 'n' =participants reporting yes for >=1 day or no for all days for specified event for each arm, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily | 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily | 13vPnC + INFANRIX Hexa
Number analyzed (Participants) | 133 | 140 | 134 | 144 | 162
percentage of participants
  Fever >=38, <=39 degree C (n= 133,140,134,144,162) | 31.6 | 37.1 | 37.3 | 50.0 | 30.2
  Fever >39, <=40 degree C (n = 128,127,118,123,150) | 5.5 | 7.1 | 4.2 | 5.7 | 2.0
  Fever >40 degree C (n = 123,125,117,122,150) | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

22. Secondary Outcome: Number of Participants With Non-Serious Adverse Events (AEs) and Serious Adverse Events (SAEs): Infant Series
Description: An AE was any untoward medical occurrence in a participant who received vaccine without regard to possibility of causal relationship. SAE: an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial/prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent events for infant series were events between infant series Dose 1 and up to 1 month (28 to 42 days) after infant series that were absent before treatment or that worsened relative to pre-treatment state. Reported non-SAEs included AEs other than SAEs collected using electronic diary (fever, systematic assessment) and events spontaneously collected on case report form at each visit (non-systematic assessment).
Time Frame: Baseline up to 1 Month (28 to 42 days) after infant series
Population: Safety analysis set Dose 1 included all participants who receive Dose 1 of 13vPnC or INFANRIX hexa in infant series and had AE or temperature data available.
Measure: Number; unit: participants
Arm/Group | 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily | 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily | 13vPnC + INFANRIX Hexa
Number analyzed (Participants) | 173 | 176 | 172 | 177 | 210
participants
  Non-SAEs | 57 | 71 | 67 | 72 | 80
  SAEs | 7 | 3 | 11 | 8 | 10

23. Secondary Outcome: Number of Participants With Non-Serious Adverse Events (AEs) and Serious Adverse Events (SAEs): After the Infant Series
Description: An AE was any untoward medical occurrence in a participant who received vaccine without regard to possibility of causal relationship. SAE: an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial/prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent events after the infant series were events between 1 month (28 to 42 days) after infant series to toddler dose that were absent before treatment or that worsened relative to pre-treatment state. Reported non-SAEs included AEs other than SAEs spontaneously collected on case report form (non-systematic assessment).
Time Frame: 1 Month (28 to 42 days) after infant series Dose 3 up to toddler dose
Population: Safety analysis set Dose 3 included all participants who receive Dose 3 of 13vPnC or INFANRIX hexa in infant series and had AE or temperature data available.
Measure: Number; unit: participants
Arm/Group | 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily | 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily | 13vPnC + INFANRIX Hexa
Number analyzed (Participants) | 170 | 174 | 172 | 176 | 210
participants
  Non-SAEs | 3 | 6 | 3 | 4 | 8
  SAEs | 6 | 14 | 10 | 11 | 9

24. Secondary Outcome: Number of Participants With Non-Serious Adverse Events (AEs) and Serious Adverse Events (SAEs): Toddler Dose
Description: An AE was any untoward medical occurrence in a participant who received vaccine without regard to possibility of causal relationship. SAE: an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial/prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent events for toddler dose were events between toddler dose and up to 1 month (28 to 42 days) after toddler dose that were absent before treatment or that worsened relative to pre-treatment state. Reported non-SAEs included AEs other than SAEs collected using electronic diary (fever, systematic assessment) and events spontaneously collected on case report form at each visit (non-systematic assessment).
Time Frame: Toddler dose up to 1 Month (28 to 42 days) after toddler dose
Population: Safety analysis set toddler dose included all participants who receive toddler dose of 13vPnC or INFANRIX hexa and had AE or temperature data available.
Measure: Number; unit: participants
Arm/Group | 13vPnC + INFANRIX Hexa + Paracetamol Twice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily | 13vPnC + INFANRIX Hexa + Paracetamol Thrice Daily | 13vPnC + INFANRIX Hexa + Ibuprofen Thrice Daily | 13vPnC + INFANRIX Hexa
Number analyzed (Participants) | 169 | 173 | 170 | 175 | 209
participants
  Non-SAEs | 47 | 57 | 52 | 76 | 50
  SAEs | 3 | 2 | 1 | 1 | 1

ADVERSE EVENTS:
Time Frame: AEs/SAEs: recorded from signing of informed consent form to completion of study. Participants recorded pre-specified AEs in electronic diary: fever (up to 4 days after each vaccine dose).
Description: Safety population: participants who received at least 1 dose of study vaccine. SAEs and AEs were grouped by system organ class and summarized. AEs included AEs collected in electronic diary (fever, systematic assessment) and events collected on case report form at each visit (nonsystematic assessment).
Groups:
- 13vPnC+ INFANRIX Hexa +Paracetamol Twice Daily -Infant Series: Participants who received 3 open-label doses (0.5 mL each) of 13vPnC intramuscularly and INFANRIX hexa intramuscularly as per manufacturer's instructions 28 to 42 days apart in infant series, along with paracetamol suspension 15 mg/kg orally at 6 to 8 hours after vaccination and 6 to 8 hours after first dose of paracetamol, assessed from Infant series Dose 1 through the blood draw 28 to 42 days post infant series.
- 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily -Infant Series: Participants who received 3 open-label doses (0.5 mL each) of 13vPnC intramuscularly and INFANRIX hexa intramuscularly as per manufacturer's instructions 28 to 42 days apart, along with ibuprofen suspension 10 mg/kg orally at 6 to 8 hours after vaccination and 6 to 8 hours after first dose of ibuprofen, assessed from Infant series Dose 1 through the blood draw 28 to 42 days post infant series.
- 13vPnC+INFANRIX Hexa+Paracetamol Thrice Daily -Infant Series: Participants who received 3 open-label doses (0.5 mL each) of 13vPnC intramuscularly and INFANRIX hexa intramuscularly as per manufacturer's instructions 28 to 42 days apart, along with paracetamol suspension 15 mg/kg orally immediately after vaccination, 6 to 8 hours after vaccination and 6 to 8 hours after last dose of paracetamol, assessed from Infant series Dose 1 through the blood draw 28 to 42 days post infant series.
- 13vPnC+ INFANRIX Hexa+ Ibuprofen Thrice Daily -Infant Series: Participants who received 3 open-label doses (0.5 mL each) of 13vPnC intramuscularly and INFANRIX hexa intramuscularly as per manufacturer's instructions 28 to 42 days apart, along with ibuprofen suspension 10 mg/kg orally immediately after vaccination, 6 to 8 hours after vaccination and 6 to 8 hours after last dose of ibuprofen, assessed from Infant series Dose 1 through the blood draw 28 to 42 days post infant series.
- 13vPnC + INFANRIX Hexa - Infant Series: Participants who received 3 open-label doses (0.5 mL each) of 13vPnC intramuscularly and INFANRIX hexa intramuscularly as per manufacturer's instructions 28 to 42 days apart, assessed from Infant series Dose 1 through the blood draw 28 to 42 days post infant series (Inf Ser).
- 13vPnC +INFANRIX Hexa +Paracetamol Twice Daily -After Inf Ser: Participants who received 3 open-label doses (0.5 mL each) of 13vPnC intramuscularly and INFANRIX hexa intramuscularly as per manufacturer's instructions 28 to 42 days apart in infant series (Inf Ser), along with paracetamol suspension 15 mg/kg orally at 6 to 8 hours after vaccination and 6 to 8 hours after first dose of paracetamol, assessed after the infant series blood draw up to toddler dose.
- 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily -After Inf Ser: Participants who received 3 open-label doses (0.5 mL each) of 13vPnC intramuscularly and INFANRIX hexa intramuscularly as per manufacturer's instructions 28 to 42 days apart in infant series (Inf Ser), along with ibuprofen suspension 10 mg/kg orally at 6 to 8 hours after vaccination and 6 to 8 hours after first dose of ibuprofen, assessed after the infant series blood draw up to toddler dose.
- 13vPnC+INFANRIX Hexa +Paracetamol Thrice Daily -After Inf Ser: Participants who received 3 open-label doses (0.5 mL each) of 13vPnC intramuscularly and INFANRIX hexa intramuscularly as per manufacturer's instructions 28 to 42 days apart in infant series (Inf Ser), along with paracetamol suspension 15 mg/kg orally immediately after vaccination, 6 to 8 hours after vaccination and 6 to 8 hours after last dose of paracetamol, assessed after the infant series blood draw up to toddler dose.
- 13vPnC +INFANRIX Hexa +Ibuprofen Thrice Daily -After Inf Ser: Participants who received 3 open-label doses (0.5 mL each) of 13vPnC intramuscularly and INFANRIX hexa intramuscularly as per manufacturer's instructions 28 to 42 days apart in infant series (Inf Ser), along with ibuprofen suspension 10 mg/kg orally immediately after vaccination, 6 to 8 hours after vaccination and 6 to 8 hours after last dose of ibuprofen, assessed after the infant series blood draw up to toddler dose.
- 13vPnC + INFANRIX Hexa - After Infant Series: Participants who received 3 open-label doses (0.5 mL each) of 13vPnC intramuscularly and INFANRIX hexa intramuscularly as per manufacturer's instructions 28 to 42 days apart in infant series, assessed after the infant series blood draw up to toddler dose.
- 13vPnC +INFANRIX Hexa + Paracetamol Twice Daily -Toddler Dose: Participants who received 3 open-label doses (0.5 mL each) of 13vPnC intramuscularly and INFANRIX hexa intramuscularly as per manufacturer's instructions 28 to 42 days apart in infant series and toddler dose (0.5 mL) of 13vPnC intramuscularly and INFANRIX hexa intramuscularly as per manufacturer's instructions at 366 to 425 days of age, along with paracetamol suspension 15 mg/kg orally at 6 to 8 hours after vaccination and 6 to 8 hours after first dose of paracetamol, assessed from the toddler dose through the blood draw 28 to 42 days post toddler dose.
- 13vPnC +INFANRIX Hexa + Ibuprofen Twice Daily -Toddler Dose: Participants who received 3 open-label doses (0.5 mL each) of 13vPnC intramuscularly and INFANRIX hexa intramuscularly as per manufacturer's instructions 28 to 42 days apart in infant series and toddler dose (0.5 mL) of 13vPnC intramuscularly and INFANRIX hexa intramuscularly as per manufacturer's instructions at 366 to 425 days of age, along with ibuprofen suspension 10 mg/kg orally at 6 to 8 hours after vaccination and 6 to 8 hours after first dose of ibuprofen, assessed from the toddler dose through the blood draw 28 to 42 days post toddler dose.
- 13vPnC +INFANRIX Hexa +Paracetamol Thrice Daily -Toddler Dose: Participants who received 3 open-label doses (0.5 mL each) of 13vPnC intramuscularly and INFANRIX hexa intramuscularly as per manufacturer's instructions 28 to 42 days apart in infant series and toddler dose (0.5 mL) of 13vPnC intramuscularly and INFANRIX hexa intramuscularly as per manufacturer's instructions at 366 to 425 days of age, along with paracetamol suspension 15 mg/kg orally immediately after vaccination, 6 to 8 hours after vaccination and 6 to 8 hours after last dose of paracetamol, assessed from the toddler dose through the blood draw 28 to 42 days post toddler dose.
- 13vPnC +INFANRIX Hexa +Ibuprofen Thrice Daily -Toddler Dose: Participants who received 3 open-label doses (0.5 mL each) of 13vPnC intramuscularly and INFANRIX hexa intramuscularly as per manufacturer's instructions 28 to 42 days apart in infant series and toddler dose (0.5 mL) of 13vPnC intramuscularly and INFANRIX hexa intramuscularly as per manufacturer's instructions at 366 to 425 days of age, along with ibuprofen suspension 15 mg/kg orally immediately after vaccination, 6 to 8 hours after vaccination and 6 to 8 hours after last dose of ibuprofen, assessed from the toddler dose through the blood draw 28 to 42 days post toddler dose.
- 13vPnC + INFANRIX Hexa - Toddler Dose: Participants who received 3 open-label doses (0.5 mL each) of 13vPnC intramuscularly and INFANRIX hexa intramuscularly as per manufacturer's instructions 28 to 42 days apart in infant series and toddler dose (0.5 mL) of 13vPnC intramuscularly and INFANRIX hexa intramuscularly as per manufacturer's instructions at 366 to 425 days of age, assessed from the toddler dose through the blood draw 28 to 42 days post toddler dose.
Arm/Group | 13vPnC+ INFANRIX Hexa +Paracetamol Twice Daily -Infant Series | 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily -Infant Series | 13vPnC+INFANRIX Hexa+Paracetamol Thrice Daily -Infant Series | 13vPnC+ INFANRIX Hexa+ Ibuprofen Thrice Daily -Infant Series | 13vPnC + INFANRIX Hexa - Infant Series | 13vPnC +INFANRIX Hexa +Paracetamol Twice Daily -After Inf Ser | 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily -After Inf Ser | 13vPnC+INFANRIX Hexa +Paracetamol Thrice Daily -After Inf Ser | 13vPnC +INFANRIX Hexa +Ibuprofen Thrice Daily -After Inf Ser | 13vPnC + INFANRIX Hexa - After Infant Series | 13vPnC +INFANRIX Hexa + Paracetamol Twice Daily -Toddler Dose | 13vPnC +INFANRIX Hexa + Ibuprofen Twice Daily -Toddler Dose | 13vPnC +INFANRIX Hexa +Paracetamol Thrice Daily -Toddler Dose | 13vPnC +INFANRIX Hexa +Ibuprofen Thrice Daily -Toddler Dose | 13vPnC + INFANRIX Hexa - Toddler Dose
Serious Adverse Events (participants affected / at risk) | 7/173 | 3/176 | 11/172 | 8/177 | 10/210 | 6/170 | 14/174 | 10/172 | 11/176 | 9/210 | 3/169 | 2/173 | 1/170 | 1/175 | 1/209
Other Adverse Events (participants affected / at risk) | 57/173 | 71/176 | 67/172 | 72/177 | 80/210 | 3/170 | 6/174 | 3/172 | 4/176 | 8/210 | 47/169 | 57/173 | 52/170 | 76/175 | 50/209
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 13vPnC+ INFANRIX Hexa +Paracetamol Twice Daily -Infant Series (N=173) | 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily -Infant Series (N=176) | 13vPnC+INFANRIX Hexa+Paracetamol Thrice Daily -Infant Series (N=172) | 13vPnC+ INFANRIX Hexa+ Ibuprofen Thrice Daily -Infant Series (N=177) | 13vPnC + INFANRIX Hexa - Infant Series (N=210) | 13vPnC +INFANRIX Hexa +Paracetamol Twice Daily -After Inf Ser (N=170) | 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily -After Inf Ser (N=174) | 13vPnC+INFANRIX Hexa +Paracetamol Thrice Daily -After Inf Ser (N=172) | 13vPnC +INFANRIX Hexa +Ibuprofen Thrice Daily -After Inf Ser (N=176) | 13vPnC + INFANRIX Hexa - After Infant Series (N=210) | 13vPnC +INFANRIX Hexa + Paracetamol Twice Daily -Toddler Dose (N=169) | 13vPnC +INFANRIX Hexa + Ibuprofen Twice Daily -Toddler Dose (N=173) | 13vPnC +INFANRIX Hexa +Paracetamol Thrice Daily -Toddler Dose (N=170) | 13vPnC +INFANRIX Hexa +Ibuprofen Thrice Daily -Toddler Dose (N=175) | 13vPnC + INFANRIX Hexa - Toddler Dose (N=209)
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 3 | 0 | 0 | 0 | 0 | 0
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Exanthema subitum (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 2 | 4 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media acute (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pertussis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 3 | 2 | 2 | 1 | 1 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 2 | 1 | 2 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis Escherichia coli (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis rotavirus (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Exposure to toxic agent (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Movement disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Breath holding (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 13vPnC+ INFANRIX Hexa +Paracetamol Twice Daily -Infant Series (N=173) | 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily -Infant Series (N=176) | 13vPnC+INFANRIX Hexa+Paracetamol Thrice Daily -Infant Series (N=172) | 13vPnC+ INFANRIX Hexa+ Ibuprofen Thrice Daily -Infant Series (N=177) | 13vPnC + INFANRIX Hexa - Infant Series (N=210) | 13vPnC +INFANRIX Hexa +Paracetamol Twice Daily -After Inf Ser (N=170) | 13vPnC + INFANRIX Hexa + Ibuprofen Twice Daily -After Inf Ser (N=174) | 13vPnC+INFANRIX Hexa +Paracetamol Thrice Daily -After Inf Ser (N=172) | 13vPnC +INFANRIX Hexa +Ibuprofen Thrice Daily -After Inf Ser (N=176) | 13vPnC + INFANRIX Hexa - After Infant Series (N=210) | 13vPnC +INFANRIX Hexa + Paracetamol Twice Daily -Toddler Dose (N=169) | 13vPnC +INFANRIX Hexa + Ibuprofen Twice Daily -Toddler Dose (N=173) | 13vPnC +INFANRIX Hexa +Paracetamol Thrice Daily -Toddler Dose (N=170) | 13vPnC +INFANRIX Hexa +Ibuprofen Thrice Daily -Toddler Dose (N=175) | 13vPnC + INFANRIX Hexa - Toddler Dose (N=209)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 1 | 3 | 7 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Dacryostenosis acquired (Eye disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 3 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 5 | 4 | 2 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 5 | 2
Dyschezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Teething (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adverse drug reaction (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Crying (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Irritability (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 6 | 5 | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 1 | 3 | 2
Vaccination site nodule (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Milk allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 9 | 8 | 11 | 9 | 5 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 3 | 5 | 2
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis infective (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Exanthema subitum (Infections and infestations) | 0 | 4 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 4 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Impetigo (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 1 | 2 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 11 | 6 | 10 | 8 | 18 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 4 | 2 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Otitis media acute (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 4 | 6 | 5 | 4 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 5 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 4 | 7 | 4 | 5 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 6 | 2
Rhinitis (Infections and infestations) | 3 | 7 | 11 | 10 | 9 | 0 | 0 | 1 | 0 | 0 | 2 | 4 | 5 | 3 | 5
Upper respiratory tract infection (Infections and infestations) | 15 | 12 | 14 | 17 | 12 | 0 | 0 | 0 | 0 | 0 | 7 | 7 | 3 | 4 | 7
Urinary tract infection (Infections and infestations) | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Varicella (Infections and infestations) | 1 | 2 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mouth injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac murmur (Investigations) | 0 | 2 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 0 | 0
Calcium metabolism disorder (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight gain poor (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertonia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotonia (Nervous system disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuromyopathy (Nervous system disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Apathy (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalciuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Genital labial adhesions (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cafe au lait spots (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 3 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 2 | 2 | 1 | 1 | 4 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin depigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Keratosis follicular (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Food allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Psychomotor retardation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vesicoureteric reflux (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast enlargement (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vaccination site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Coxsackie viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fever >=38, <=39 degree C (General disorders) | 49/149 | 71/157 | 27/147 | 53/155 | 78/187 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 42/133 | 52/140 | 50/134 | 72/144 | 49/162 — Infant Series Dose 1 and Toddler Dose
Fever >39, <=40 degree C (General disorders) | 2/138 | 2/145 | 1/137 | 1/146 | 2/170 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 7/128 | 9/127 | 5/118 | 7/123 | 3/150 — Infant Series Dose 1 and Toddler Dose
Fever >40 degree C (General disorders) | 0/138 | 0/145 | 0/137 | 0/146 | 0/170 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/123 | 0/125 | 0/117 | 0/122 | 0/150 — Infant Series Dose 1 and Toddler Dose
Fever >=38, <=39 degree C (General disorders) | 37/141 | 65/152 | 30/140 | 70/159 | 72/181 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2
Fever >39, <=40 degree C (General disorders) | 2/133 | 1/140 | 2/134 | 2/145 | 6/164 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2
Fever >40 degree C (General disorders) | 0/131 | 0/140 | 0/133 | 0/144 | 0/164 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2
Fever >=38, <=39 degree C (General disorders) | 30/136 | 45/146 | 23/135 | 47/141 | 52/175 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3
Fever >39, <=40 degree C (General disorders) | 2/129 | 4/137 | 1/125 | 2/136 | 3/167 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3
Fever >40 degree C (General disorders) | 0/128 | 0/136 | 1/126 | 0/135 | 0/166 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3. Report of fever >40 degrees C after 13vPnC Infant Series Dose 3 was confirmed as data entry error.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.